CLINICAL TRIAL: NCT02531698
Title: A Phase 2, Randomized, Controlled, Observer-blinded Study To Describe The Immunogenicity, Safety, And Tolerability Of Neisseria Meningitidis Serogroup B Bivalent Recombinant Lipoprotein 2086 Vaccine (Bivalent Rlp2086) In Healthy Subjects Aged >/= 24 Months To <10 Years
Brief Title: A Study to Describe the Immunogenicity, Safety, and Tolerability of Neisseria Meningitidis Serogroup B Bivalent Recombinant Lipoprotein 2086 Vaccine (Bivalent rLP2086) in Healthy Subjects Aged ≥24 Months to <10 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B1971017; 2014-000933-21 (EudraCT Number); 6108K2-3012 (Other: Alias Study Number)
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: MENINGOCOCCAL INFECTION
MeSH Terms: conditions — Meningococcal Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bivalent rLP2086 (Experimental): Bivalent rLP2086 (containing 60 μg each of a purified subfamily A and subfamily B rLP2086 protein, adsorbed to aluminum in a sterile buffered isotonic suspension) in a 0.5-mL dose for injection.
  Interventions: Biological: Bivalent rLP2086 Vaccine
- Licensed pediatric hepatitis A vaccine (Other)
  Interventions: Biological: Licensed pediatric hepatits A vaccine; Other: Normal Saline

INTERVENTIONS:
Biological: Bivalent rLP2086 Vaccine — 1 dose of 120 μg of bivalent rLP2086 by intramuscular injection at Months 0, 2, and 6 into the upper deltoid muscle of the arm.
  Arms: Bivalent rLP2086
Biological: Licensed pediatric hepatits A vaccine — 1 0.5 mL dose by intramuscular injection at Months 0 and 6 into the upper deltoid muscle of the arm.
  Arms: Licensed pediatric hepatitis A vaccine
Other: Normal Saline — Sterile saline solution for injection (0.85% sodium chloride) in a 0.5 mL dose at Month 2.
  Arms: Licensed pediatric hepatitis A vaccine

SUMMARY:
This study is looking at a new vaccine that might prevent meningococcal disease, and will study the immune response elicited by this vaccine when given to healthy young children. The study will also look at the safety of the new vaccine as well as how it is tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document (ICD) indicating that the subject's parent(s)/legal guardian has been informed of all pertinent aspects of the study.
2. Parent(s)/legal guardian and subject who are willing and able to comply with scheduled visits, vaccine regimen, laboratory tests, and other study procedures.
3. Male or female subjects aged ≥24 months and <10 years at time of randomization, stratified equally by age (≥24 months to <4 years or ≥4 years to <10 years).
4. Subject is available for the entire study period and subject's parent(s)/legal guardian can be reached by telephone.
5. Healthy subject as determined by medical history, physical examination, and judgment of the investigator.
6. Subject must have received all vaccinations in the relevant national immunization program (NIP) for their age group.
7. Male and female subjects of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study. A subject is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active.
8. Negative urine pregnancy test for all female subjects who are biologically capable of having children.

Exclusion Criteria:

1. Previous vaccination with any meningococcal serogroup B vaccine.
2. Subjects who have received prior HAV vaccination.
3. Contraindication to vaccination with any HAV vaccine or known latex allergy.
4. Subjects receiving any allergen immunotherapy with a nonlicensed product or subjects receiving allergen immunotherapy with a licensed product and who are not on stable maintenance doses.
5. A previous anaphylactic reaction to any vaccine or vaccine-related component.
6. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
7. A known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as subjects with congenital or acquired defects in B-cell function, those receiving chronic systemic (oral, intravenous, or intramuscular) corticosteroid therapy, or those receiving immunosuppressive therapy. Subjects with terminal complement deficiency may be included. Additional details will be provided in the study reference manual (SRM).
8. History of microbiologically proven disease caused by N meningitidis or Neisseria gonorrhoeae.
9. Significant neurological disorder or history of seizure (excluding simple febrile seizure).
10. Receipt of any blood products, including immunoglobulin, within 6 months before the first study vaccination.
11. Current chronic use of systemic antibiotics.
12. Participation in other studies involving investigational product(s)/device(s) (Phases 1-4) within 28 days before administration of the first study vaccination. Participation in purely observational studies is acceptable.
13. Any neuroinflammatory or autoimmune condition, including but not limited to transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.
14. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
15. Pregnant female subjects, breastfeeding female subjects, male subjects with partners who are currently pregnant, or male and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study.
16. Subjects who are children of investigational site staff members directly involved in the conduct of the study and their family members, subjects who are children of site staff members otherwise supervised by the investigator, or subjects who are children of Pfizer employees directly involved in the conduct of the study.

Ages: 24 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- Finland (7):
  - Espoo Vaccine Research Clinic, Espoo
  - Helsinki South Vaccine Research Clinic, Helsinki
  - Oulu Vaccine Research Clinic, Oulu
  - Pori Vaccine Research Clinic, Pori
  - Tampere Vaccine Research Clinic, Tampere
  - Turku Vaccine Research Center, Turku
  - Turku Vaccine Research Clinic, Turku
- Poland (8):
  - Prywatny Gabinet Lekarski dr n. med. Jerzy Brzostek, Dębica
  - Praktyka Lekarza Rodzinnego-Slawin Sp. z o.o., Kiełczów
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Hanna Czajka - Indywidualna Specjalistyczna Praktyka Lekarska, Krakow
  - Specjalistyczna Przychodnia Medycyny Wieku Rozwojowego, Poznan
  - Niepubliczny Zaklad Lecznictwa Ambulatoryjnego "Michalkowice"Jarosz i Partnerzy Spolka Lekarska, Siemianowice Śląskie
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 We Wroclawiu, Wroclaw
  - Niepubliczny Zaklad Opieki Zdrowotnej Salmed S. C., Łęczna

REFERENCES:
- [Derived] Marshall HS, Vesikari T, Richmond PC, Wysocki J, Szenborn L, Beeslaar J, Maguire JD, Balmer P, O'Neill R, Anderson AS, Pregaldien JL, Maansson R, Jiang HQ, Perez JL. Safety and immunogenicity of a primary series and booster dose of the meningococcal serogroup B-factor H binding protein vaccine (MenB-FHbp) in healthy children aged 1-9 years: two phase 2 randomised, controlled, observer-blinded studies. Lancet Infect Dis. 2023 Jan;23(1):103-116. doi: 10.1016/S1473-3099(22)00424-8. Epub 2022 Sep 7. PMID 36087588
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1971017&StudyName=A%20Phase%202%2C%20Randomized%2C%20Controlled%2C%20Observer-blinded%20Study%20To%20Describe%20The%20Immunogenicity%2C%20Safety%2C%20And%20Tolerability%20Of%20Neisseria%20Meningitidis%20Serogroup%20B%20Bivalent%20Recombinant%20Lipoprotein%202086%20Vaccine%20%28bivalent%20Rlp2086%29%20In%20Healthy%20Subjects%20Aged%20greater%20than%2F%3D%2024%20Months%20To%20less%20than10%20Years

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Bivalent rLP2086 (>=24 Months to <10 Years): Participants from greater than or equal to (>=) 24 months to less than (<) 10 years of age, received intramuscular injection of rLP2086 vaccine on a 0-, 2-, 6- month schedule.
- Group 2 HAV/Saline (>=24 Months to <10 Years): Participants from >=24 months to <10 years of age, received intramuscular injection of saline on 2- month and HAV vaccine on a 0-, 6- month schedule.
Period: Overall Study
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years)
Started | 294 | 106
Completed | 283 | 104
Not Completed | 11 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of the investigational product (rLP2086, HAV vaccine or saline) and had safety data available.
Groups:
- Group 1 Bivalent rLP2086 (>=24 Months to <10 Years): Participants from >=24 months to <10 years of age, received intramuscular injection of rLP2086 vaccine on a 0-, 2-, 6- month schedule.
- Total: Total of all reporting groups
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Total
Number analyzed (Participants) | 294 | 106 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.3 (2.24) | 4.2 (2.15) | 4.3 (2.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 62 | 208
  Male | 148 | 44 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 294 | 106 | 400
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 291 | 104 | 395
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titers >= Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Neisseria Meningitidis Serogroup B (MnB) Test Strains 1 Month After Vaccination 3
Description: Percentage of participants achieving hSBA titer >= LLOQ were computed along with corresponding 2-sided 95 percent (%) confidence interval (CIs). LLOQ was 1:16 for PMB80 (A22) and 1:8 for PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44).
Time Frame: 1 month after Vaccination 3
Population: Evaluable immunogenicity population: all eligible participants randomized to study, received scheduled investigational products, had pre and post vaccination blood drawn with valid and determinate assay results and had no important protocol deviation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Group 1 Bivalent rLP2086 (>=24 Months to <4 Years): Participants from >=24 months to <4 years of age, received intramuscular injection of rLP2086 vaccine on a 0-, 2-, 6- month schedule.
- Group 1 Bivalent rLP2086 (>=4 Years to <10 Years): Participants from >=4 years to <10 years of age, received intramuscular injection of rLP2086 vaccine on a 0-, 2-, 6- month schedule.
- Group 2 HAV/Saline (>=24 Months to <4 Years): Participants from >=24 months to <4 years of age, received intramuscular injection of saline on 2- month and HAV vaccine on a 0-, 6- month schedule.
- Group 2 HAV/Saline (>=4 Years to <10 Years): Participants from >=4 years to <10 years of age, received intramuscular injection of saline on 2- month and HAV vaccine on a 0-, 6- month schedule.
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 136 | 138 | 52 | 45
Percentage of participants
  PMB80 [A22]: number analyzed (Participants) | 68 | 67 | 25 | 20
  PMB80 [A22] | 83.8 [72.9 to 91.6] | 91.0 [81.5 to 96.6] | 4.0 [0.1 to 20.4] | 10.0 [1.2 to 31.7]
  PMB2001 [A56]: number analyzed (Participants) | 68 | 71 | 24 | 19
  PMB2001 [A56] | 100.0 [94.7 to 100.0] | 100.0 [94.9 to 100.0] | 4.2 [0.1 to 21.1] | 42.1 [20.3 to 66.5]
  PMB2948 [B24]: number analyzed (Participants) | 63 | 63 | 26 | 20
  PMB2948 [B24] | 85.7 [74.6 to 93.3] | 92.1 [82.4 to 97.4] | 7.7 [0.9 to 25.1] | 0.0 [0.0 to 16.8]
  PMB2707 [B44]: number analyzed (Participants) | 65 | 69 | 26 | 24
  PMB2707 [B44] | 80.0 [68.2 to 88.9] | 78.3 [66.7 to 87.3] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]

2. Primary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 7 Days After Vaccination 1
Description: Local reactions included pain at injection site, swelling and redness collected by using an electronic diary (e-diary). Pain was graded as: mild (did not interfere with activity), moderate (interfered with activity) and severe (prevented daily activity). Redness and swelling were graded as: mild (0.5-2.0 centimeter [cm]), moderate (2.5 to 7.0 cm) and severe (>7.0 cm).
Time Frame: Within 7 Days after Vaccination 1
Population: Vaccination 1 safety population: all participants who received the first dose of investigational products (rLP2086 or HAV vaccine) on Day 1 (Month 0).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants
  Pain at injection site: Any | 66.0 [60.3 to 71.4] | 51.7 [43.3 to 60.1] | 79.9 [72.5 to 86.0] | 22.6 [15.1 to 31.8] | 10.9 [4.1 to 22.2] | 35.3 [22.4 to 49.9]
  Pain at injection site: Mild | 32.3 [27.0 to 38.0] | 24.1 [17.4 to 31.9] | 40.3 [32.3 to 48.6] | 17.9 [11.2 to 26.6] | 9.1 [3.0 to 20.0] | 27.5 [15.9 to 41.7]
  Pain at injection site: Moderate | 30.3 [25.1 to 35.9] | 24.8 [18.0 to 32.7] | 35.6 [27.9 to 43.8] | 4.7 [1.5 to 10.7] | 1.8 [0.0 to 9.7] | 7.8 [2.2 to 18.9]
  Pain at injection site: Severe | 3.4 [1.6 to 6.2] | 2.8 [0.8 to 6.9] | 4.0 [1.5 to 8.6] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]
  Redness: Any | 40.8 [35.1 to 46.7] | 42.1 [33.9 to 50.5] | 39.6 [31.7 to 47.9] | 9.4 [4.6 to 16.7] | 10.9 [4.1 to 22.2] | 7.8 [2.2 to 18.9]
  Redness: Mild | 17.7 [13.5 to 22.5] | 22.1 [15.6 to 29.7] | 13.4 [8.4 to 20.0] | 5.7 [2.1 to 11.9] | 7.3 [2.0 to 17.6] | 3.9 [0.5 to 13.5]
  Redness: Moderate | 18.7 [14.4 to 23.6] | 18.6 [12.6 to 25.9] | 18.8 [12.9 to 26.0] | 3.8 [1.0 to 9.4] | 3.6 [0.4 to 12.5] | 3.9 [0.5 to 13.5]
  Redness: Severe | 4.4 [2.4 to 7.4] | 1.4 [0.2 to 4.9] | 7.4 [3.7 to 12.8] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]
  Swelling: Any | 31.3 [26.0 to 36.9] | 27.6 [20.5 to 35.6] | 34.9 [27.3 to 43.1] | 5.7 [2.1 to 11.9] | 5.5 [1.1 to 15.1] | 5.9 [1.2 to 16.2]
  Swelling: Mild | 12.2 [8.7 to 16.5] | 11.0 [6.4 to 17.3] | 13.4 [8.4 to 20.0] | 3.8 [1.0 to 9.4] | 3.6 [0.4 to 12.5] | 3.9 [0.5 to 13.5]
  Swelling: Moderate | 17.3 [13.2 to 22.2] | 16.6 [10.9 to 23.6] | 18.1 [12.3 to 25.3] | 1.9 [0.2 to 6.6] | 1.8 [0.0 to 9.7] | 2.0 [0.0 to 10.4]
  Swelling: Severe | 1.7 [0.6 to 3.9] | 0.0 [0.0 to 2.5] | 3.4 [1.1 to 7.7] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]

3. Primary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 7 Days After Vaccination 2
Description: Local reactions included pain at injection site, swelling and redness collected by using an e-diary. Pain was graded as: mild (did not interfere with activity), moderate (interfered with activity) and severe (prevented daily activity). Redness and swelling were graded as: mild (0.5-2.0 cm), moderate (2.5 to 7.0 cm) and severe (>7.0 cm).
Time Frame: Within 7 Days after Vaccination 2
Population: Vaccination 2 safety population: all participants who received the second dose of investigational products (rLP2086 or saline) on Month 2 visit. Here "number of participants analyzed (N)" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 291 | 143 | 148 | 103 | 54 | 49
Percentage of participants
  Pain at injection site: Any | 70.8 [65.2 to 76.0] | 63.6 [55.2 to 71.5] | 77.7 [70.1 to 84.1] | 12.6 [6.9 to 20.6] | 5.6 [1.2 to 15.4] | 20.4 [10.2 to 34.3]
  Pain at injection site: Mild | 40.2 [34.5 to 46.1] | 40.6 [32.4 to 49.1] | 39.9 [31.9 to 48.2] | 9.7 [4.8 to 17.1] | 5.6 [1.2 to 15.4] | 14.3 [5.9 to 27.2]
  Pain at injection site: Moderate | 28.5 [23.4 to 34.1] | 20.3 [14.0 to 27.8] | 36.5 [28.7 to 44.8] | 2.9 [0.6 to 8.3] | 0.0 [0.0 to 6.6] | 6.1 [1.3 to 16.9]
  Pain at injection site: Severe | 2.1 [0.8 to 4.4] | 2.8 [0.8 to 7.0] | 1.4 [0.2 to 4.8] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Redness: Any | 37.1 [31.5 to 42.9] | 36.4 [28.5 to 44.8] | 37.8 [30.0 to 46.2] | 5.8 [2.2 to 12.2] | 5.6 [1.2 to 15.4] | 6.1 [1.3 to 16.9]
  Redness: Mild | 16.5 [12.4 to 21.3] | 15.4 [9.9 to 22.4] | 17.6 [11.8 to 24.7] | 5.8 [2.2 to 12.2] | 5.6 [1.2 to 15.4] | 6.1 [1.3 to 16.9]
  Redness: Moderate | 18.2 [14.0 to 23.1] | 20.3 [14.0 to 27.8] | 16.2 [10.7 to 23.2] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Redness: Severe | 2.4 [1.0 to 4.9] | 0.7 [0.0 to 3.8] | 4.1 [1.5 to 8.6] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Swelling: Any | 28.5 [23.4 to 34.1] | 27.3 [20.2 to 35.3] | 29.7 [22.5 to 37.8] | 1.0 [0.0 to 5.3] | 0.0 [0.0 to 6.6] | 2.0 [0.1 to 10.9]
  Swelling: Mild | 11.7 [8.2 to 15.9] | 11.9 [7.1 to 18.4] | 11.5 [6.8 to 17.8] | 1.0 [0.0 to 5.3] | 0.0 [0.0 to 6.6] | 2.0 [0.1 to 10.9]
  Swelling: Moderate | 16.2 [12.1 to 20.9] | 14.7 [9.3 to 21.6] | 17.6 [11.8 to 24.7] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Swelling: Severe | 0.7 [0.1 to 2.5] | 0.7 [0.0 to 3.8] | 0.7 [0.0 to 3.7] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]

4. Primary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 7 Days After Vaccination 3
Description: as for outcome 3
Time Frame: Within 7 Days after Vaccination 3
Population: Vaccination 3 safety population: all participants who received the third dose of investigational product (rLP2086 or HAV vaccine) on Month 6 visit. Here "N" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 285 | 139 | 146 | 104 | 54 | 50
Percentage of participants
  Pain at injection site: Any | 68.4 [62.7 to 73.8] | 54.7 [46.0 to 63.1] | 81.5 [74.2 to 87.4] | 15.4 [9.1 to 23.8] | 9.3 [3.1 to 20.3] | 22.0 [11.5 to 36.0]
  Pain at injection site: Mild | 38.2 [32.6 to 44.2] | 26.6 [19.5 to 34.8] | 49.3 [41.0 to 57.7] | 10.6 [5.4 to 18.1] | 7.4 [2.1 to 17.9] | 14.0 [5.8 to 26.7]
  Pain at injection site: Moderate | 27.0 [21.9 to 32.6] | 25.2 [18.2 to 33.2] | 28.8 [21.6 to 36.8] | 4.8 [1.6 to 10.9] | 1.9 [0.0 to 9.9] | 8.0 [2.2 to 19.2]
  Pain at injection site: Severe | 3.2 [1.5 to 5.9] | 2.9 [0.8 to 7.2] | 3.4 [1.1 to 7.8] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]
  Redness: Any | 35.1 [29.6 to 40.9] | 34.5 [26.7 to 43.1] | 35.6 [27.9 to 44.0] | 9.6 [4.7 to 17.0] | 9.3 [3.1 to 20.3] | 10.0 [3.3 to 21.8]
  Redness: Mild | 16.5 [12.4 to 21.3] | 15.8 [10.2 to 23.0] | 17.1 [11.4 to 24.2] | 8.7 [4.0 to 15.8] | 7.4 [2.1 to 17.9] | 10.0 [3.3 to 21.8]
  Redness: Moderate | 14.7 [10.8 to 19.4] | 17.3 [11.4 to 24.6] | 12.3 [7.5 to 18.8] | 1.0 [0.0 to 5.2] | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 7.1]
  Redness: Severe | 3.9 [1.9 to 6.8] | 1.4 [0.2 to 5.1] | 6.2 [2.9 to 11.4] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]
  Swelling: Any | 27.4 [22.3 to 32.9] | 24.5 [17.6 to 32.5] | 30.1 [22.8 to 38.3] | 4.8 [1.6 to 10.9] | 3.7 [0.5 to 12.7] | 6.0 [1.3 to 16.5]
  Swelling: Mild | 11.9 [8.4 to 16.3] | 9.4 [5.1 to 15.5] | 14.4 [9.1 to 21.1] | 3.8 [1.1 to 9.6] | 1.9 [0.0 to 9.9] | 6.0 [1.3 to 16.5]
  Swelling: Moderate | 14.7 [10.8 to 19.4] | 15.1 [9.6 to 22.2] | 14.4 [9.1 to 21.1] | 1.0 [0.0 to 5.2] | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 7.1]
  Swelling: Severe | 0.7 [0.1 to 2.5] | 0.0 [0.0 to 2.6] | 1.4 [0.2 to 4.9] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]

5. Primary Outcome: Percentage of Participants Reporting Systemic Events and Antipyretic Use Within 7 Days After Vaccination 1
Description: Systemic reactions included fever, vomiting, diarrhea, headache, fatigue, muscle and joint pain (other than at the injection site) and recorded by using an e-diary. Fever was graded as 38.0 to 38.4 degree Celsius (C), 38.5 to 38.9 degree C, 39.0 to 39.4 degree C, >39.5 to 40.0 degree C and >40.0 degree C. Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours) and severe (required intravenous hydration). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours) and severe (>=6 loose stools in 24 hours). Headache, fatigue, muscle pain and joint pain were graded as mild (no interference with activity), moderate (some interference with activity) and severe (prevented daily activity).
Time Frame: Within 7 Days after Vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants
  Fever >=38 degrees C | 16.3 [12.3 to 21.1] | 21.4 [15.0 to 29.0] | 11.4 [6.8 to 17.6] | 6.6 [2.7 to 13.1] | 10.9 [4.1 to 22.2] | 2.0 [0.0 to 10.4]
  Fever 38 to <38.5 degrees C | 6.1 [3.7 to 9.5] | 6.9 [3.4 to 12.3] | 5.4 [2.3 to 10.3] | 4.7 [1.5 to 10.7] | 7.3 [2.0 to 17.6] | 2.0 [0.0 to 10.4]
  Fever 38.5 to <39 degrees C | 6.1 [3.7 to 9.5] | 7.6 [3.8 to 13.2] | 4.7 [1.9 to 9.4] | 1.9 [0.2 to 6.6] | 3.6 [0.4 to 12.5] | 0.0 [0.0 to 7.0]
  Fever 39 to <39.5 degrees C | 2.4 [1.0 to 4.8] | 3.4 [1.1 to 7.9] | 1.3 [0.2 to 4.8] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]
  Fever 39.5 to 40 degrees C | 1.4 [0.4 to 3.4] | 2.8 [0.8 to 6.9] | 0.0 [0.0 to 2.4] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]
  Fever >40 degrees C | 0.3 [0.0 to 1.9] | 0.7 [0.0 to 3.8] | 0.0 [0.0 to 2.4] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]
  Vomiting: Any | 5.4 [3.1 to 8.7] | 9.0 [4.9 to 14.8] | 2.0 [0.4 to 5.8] | 3.8 [1.0 to 9.4] | 5.5 [1.1 to 15.1] | 2.0 [0.0 to 10.4]
  Vomiting: Mild | 4.4 [2.4 to 7.4] | 7.6 [3.8 to 13.2] | 1.3 [0.2 to 4.8] | 2.8 [0.6 to 8.0] | 5.5 [1.1 to 15.1] | 0.0 [0.0 to 7.0]
  Vomiting: Moderate | 1.0 [0.2 to 3.0] | 1.4 [0.2 to 4.9] | 0.7 [0.0 to 3.7] | 0.9 [0.0 to 5.1] | 0.0 [0.0 to 6.5] | 2.0 [0.0 to 10.4]
  Vomiting: Severe | 0.0 [0.0 to 1.2] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 2.4] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]
  Diarrhea: Any | 9.2 [6.1 to 13.1] | 11.7 [7.0 to 18.1] | 6.7 [3.3 to 12.0] | 6.6 [2.7 to 13.1] | 7.3 [2.0 to 17.6] | 5.9 [1.2 to 16.2]
  Diarrhea: Mild | 7.1 [4.5 to 10.7] | 9.0 [4.9 to 14.8] | 5.4 [2.3 to 10.3] | 6.6 [2.7 to 13.1] | 7.3 [2.0 to 17.6] | 5.9 [1.2 to 16.2]
  Diarrhea: Moderate | 1.7 [0.6 to 3.9] | 2.1 [0.4 to 5.9] | 1.3 [0.2 to 4.8] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]
  Diarrhea: Severe | 0.3 [0.0 to 1.9] | 0.7 [0.0 to 3.8] | 0.0 [0.0 to 2.4] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]
  Headache: Any | 18.4 [14.1 to 23.3] | 8.3 [4.3 to 14.0] | 28.2 [21.1 to 36.1] | 11.3 [6.0 to 18.9] | 3.6 [0.4 to 12.5] | 19.6 [9.8 to 33.1]
  Headache: Mild | 9.5 [6.4 to 13.5] | 3.4 [1.1 to 7.9] | 15.4 [10.0 to 22.3] | 6.6 [2.7 to 13.1] | 1.8 [0.0 to 9.7] | 11.8 [4.4 to 23.9]
  Headache: Moderate | 8.5 [5.6 to 12.3] | 4.8 [2.0 to 9.7] | 12.1 [7.3 to 18.4] | 3.8 [1.0 to 9.4] | 1.8 [0.0 to 9.7] | 5.9 [1.2 to 16.2]
  Headache: Severe | 0.3 [0.0 to 1.9] | 0.0 [0.0 to 2.5] | 0.7 [0.0 to 3.7] | 0.9 [0.0 to 5.1] | 0.0 [0.0 to 6.5] | 2.0 [0.0 to 10.4]
  Fatigue: Any | 49.0 [43.1 to 54.8] | 55.9 [47.4 to 64.1] | 42.3 [34.2 to 50.6] | 25.5 [17.5 to 34.9] | 20.0 [10.4 to 33.0] | 31.4 [19.1 to 45.9]
  Fatigue: Mild | 21.8 [17.2 to 26.9] | 24.1 [17.4 to 31.9] | 19.5 [13.4 to 26.7] | 14.2 [8.1 to 22.3] | 9.1 [3.0 to 20.0] | 19.6 [9.8 to 33.1]
  Fatigue: Moderate | 23.5 [18.7 to 28.7] | 27.6 [20.5 to 35.6] | 19.5 [13.4 to 26.7] | 8.5 [4.0 to 15.5] | 5.5 [1.1 to 15.1] | 11.8 [4.4 to 23.9]
  Fatigue: Severe | 3.7 [1.9 to 6.6] | 4.1 [1.5 to 8.8] | 3.4 [1.1 to 7.7] | 2.8 [0.6 to 8.0] | 5.5 [1.1 to 15.1] | 0.0 [0.0 to 7.0]
  Muscle pain : Any | 16.3 [12.3 to 21.1] | 13.1 [8.1 to 19.7] | 19.5 [13.4 to 26.7] | 5.7 [2.1 to 11.9] | 1.8 [0.0 to 9.7] | 9.8 [3.3 to 21.4]
  Muscle pain : Mild | 8.8 [5.9 to 12.7] | 6.2 [2.9 to 11.5] | 11.4 [6.8 to 17.6] | 4.7 [1.5 to 10.7] | 1.8 [0.0 to 9.7] | 7.8 [2.2 to 18.9]
  Muscle pain : Moderate | 6.1 [3.7 to 9.5] | 4.8 [2.0 to 9.7] | 7.4 [3.7 to 12.8] | 0.9 [0.0 to 5.1] | 0.0 [0.0 to 6.5] | 2.0 [0.0 to 10.4]
  Muscle pain : Severe | 1.4 [0.4 to 3.4] | 2.1 [0.4 to 5.9] | 0.7 [0.0 to 3.7] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]
  Joint pain: Any | 6.5 [3.9 to 9.9] | 6.2 [2.9 to 11.5] | 6.7 [3.3 to 12.0] | 4.7 [1.5 to 10.7] | 1.8 [0.0 to 9.7] | 7.8 [2.2 to 18.9]
  Joint pain: Mild | 3.4 [1.6 to 6.2] | 3.4 [1.1 to 7.9] | 3.4 [1.1 to 7.7] | 4.7 [1.5 to 10.7] | 1.8 [0.0 to 9.7] | 7.8 [2.2 to 18.9]
  Joint pain: Moderate | 3.1 [1.4 to 5.7] | 2.8 [0.8 to 6.9] | 3.4 [1.1 to 7.7] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]
  Joint pain: Severe | 0.0 [0.0 to 1.2] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 2.4] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]
  Antipyretic Medication Use | 37.1 [31.5 to 42.9] | 42.8 [34.6 to 51.2] | 31.5 [24.2 to 39.7] | 16.0 [9.6 to 24.4] | 14.5 [6.5 to 26.7] | 17.6 [8.4 to 30.9]

6. Primary Outcome: Percentage of Participants Reporting Systemic Events and Antipyretic Use Within 7 Days After Vaccination 2
Description: Systemic reactions included fever, vomiting, diarrhea, headache, fatigue, muscle and joint pain (other than at the injection site) and recorded by using an e-diary. Fever was graded as 38.0 to 38.4 degree C, 38.5 to 38.9 degree C, 39.0 to 39.4 degree C, >39.5 to 40.0 degree C and >40.0 degree C. Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours) and severe (required intravenous hydration). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours) and severe (>=6 loose stools in 24 hours). Headache, fatigue, muscle pain and joint pain were graded as mild (no interference with activity), moderate (some interference with activity) and severe (prevented daily activity).
Time Frame: Within 7 Days after Vaccination 2
Population: Vaccination 2 safety population: all participants who received the second dose of investigational products (rLP2086 or saline) on Month 2 visit. Here "N" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 291 | 143 | 148 | 103 | 54 | 49
Percentage of participants
  Fever >=38 degrees C | 12.0 [8.5 to 16.3] | 15.4 [9.9 to 22.4] | 8.8 [4.8 to 14.6] | 2.9 [0.6 to 8.3] | 3.7 [0.5 to 12.7] | 2.0 [0.1 to 10.9]
  Fever 38 to <38.5 degrees C | 6.5 [4.0 to 10.0] | 7.7 [3.9 to 13.3] | 5.4 [2.4 to 10.4] | 1.9 [0.2 to 6.8] | 3.7 [0.5 to 12.7] | 0.0 [0.0 to 7.3]
  Fever 38.5 to <39 degrees C | 1.7 [0.6 to 4.0] | 2.8 [0.8 to 7.0] | 0.7 [0.0 to 3.7] | 1.0 [0.0 to 5.3] | 0.0 [0.0 to 6.6] | 2.0 [0.1 to 10.9]
  Fever 39 to <39.5 degrees C | 1.7 [0.6 to 4.0] | 1.4 [0.2 to 5.0] | 2.0 [0.4 to 5.8] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Fever 39.5 to 40 degrees C | 1.7 [0.6 to 4.0] | 2.8 [0.8 to 7.0] | 0.7 [0.0 to 3.7] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Fever >40 degrees C | 0.3 [0.0 to 1.9] | 0.7 [0.0 to 3.8] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Vomiting: Any | 5.2 [2.9 to 8.4] | 5.6 [2.4 to 10.7] | 4.7 [1.9 to 9.5] | 4.9 [1.6 to 11.0] | 3.7 [0.5 to 12.7] | 6.1 [1.3 to 16.9]
  Vomiting: Mild | 3.4 [1.7 to 6.2] | 4.2 [1.6 to 8.9] | 2.7 [0.7 to 6.8] | 3.9 [1.1 to 9.6] | 1.9 [0.0 to 9.9] | 6.1 [1.3 to 16.9]
  Vomiting: Moderate | 1.7 [0.6 to 4.0] | 1.4 [0.2 to 5.0] | 2.0 [0.4 to 5.8] | 1.0 [0.0 to 5.3] | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 7.3]
  Vomiting: Severe | 0.0 [0.0 to 1.3] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Diarrhea: Any | 8.2 [5.4 to 12.0] | 9.8 [5.5 to 15.9] | 6.8 [3.3 to 12.1] | 5.8 [2.2 to 12.2] | 5.6 [1.2 to 15.4] | 6.1 [1.3 to 16.9]
  Diarrhea: Mild | 7.6 [4.8 to 11.2] | 8.4 [4.4 to 14.2] | 6.8 [3.3 to 12.1] | 5.8 [2.2 to 12.2] | 5.6 [1.2 to 15.4] | 6.1 [1.3 to 16.9]
  Diarrhea: Moderate | 0.3 [0.0 to 1.9] | 0.7 [0.0 to 3.8] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Diarrhea: Severe | 0.3 [0.0 to 1.9] | 0.7 [0.0 to 3.8] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Headache: Any | 18.2 [14.0 to 23.1] | 11.2 [6.5 to 17.5] | 25.0 [18.3 to 32.8] | 11.7 [6.2 to 19.5] | 1.9 [0.0 to 9.9] | 22.4 [11.8 to 36.6]
  Headache: Mild | 10.3 [7.1 to 14.4] | 7.7 [3.9 to 13.3] | 12.8 [7.9 to 19.3] | 9.7 [4.8 to 17.1] | 1.9 [0.0 to 9.9] | 18.4 [8.8 to 32.0]
  Headache: Moderate | 7.6 [4.8 to 11.2] | 3.5 [1.1 to 8.0] | 11.5 [6.8 to 17.8] | 1.0 [0.0 to 5.3] | 0.0 [0.0 to 6.6] | 2.0 [0.1 to 10.9]
  Headache: Severe | 0.3 [0.0 to 1.9] | 0.0 [0.0 to 2.5] | 0.7 [0.0 to 3.7] | 1.0 [0.0 to 5.3] | 0.0 [0.0 to 6.6] | 2.0 [0.1 to 10.9]
  Fatigue: Any | 43.3 [37.5 to 49.2] | 45.5 [37.1 to 54.0] | 41.2 [33.2 to 49.6] | 13.6 [7.6 to 21.8] | 13.0 [5.4 to 24.9] | 14.3 [5.9 to 27.2]
  Fatigue: Mild | 21.0 [16.4 to 26.1] | 22.4 [15.8 to 30.1] | 19.6 [13.5 to 26.9] | 7.8 [3.4 to 14.7] | 7.4 [2.1 to 17.9] | 8.2 [2.3 to 19.6]
  Fatigue: Moderate | 19.6 [15.2 to 24.6] | 19.6 [13.4 to 27.0] | 19.6 [13.5 to 26.9] | 5.8 [2.2 to 12.2] | 5.6 [1.2 to 15.4] | 6.1 [1.3 to 16.9]
  Fatigue: Severe | 2.7 [1.2 to 5.3] | 3.5 [1.1 to 8.0] | 2.0 [0.4 to 5.8] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Muscle pain: Any | 13.1 [9.4 to 17.5] | 11.2 [6.5 to 17.5] | 14.9 [9.6 to 21.6] | 1.9 [0.2 to 6.8] | 0.0 [0.0 to 6.6] | 4.1 [0.5 to 14.0]
  Muscle pain: Mild | 6.9 [4.2 to 10.4] | 3.5 [1.1 to 8.0] | 10.1 [5.8 to 16.2] | 1.9 [0.2 to 6.8] | 0.0 [0.0 to 6.6] | 4.1 [0.5 to 14.0]
  Muscle pain: Moderate | 5.8 [3.4 to 9.2] | 7.0 [3.4 to 12.5] | 4.7 [1.9 to 9.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Muscle pain: Severe | 0.3 [0.0 to 1.9] | 0.7 [0.0 to 3.8] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Joint pain: Any | 7.2 [4.5 to 10.8] | 5.6 [2.4 to 10.7] | 8.8 [4.8 to 14.6] | 3.9 [1.1 to 9.6] | 0.0 [0.0 to 6.6] | 8.2 [2.3 to 19.6]
  Joint pain: Mild | 2.7 [1.2 to 5.3] | 1.4 [0.2 to 5.0] | 4.1 [1.5 to 8.6] | 3.9 [1.1 to 9.6] | 0.0 [0.0 to 6.6] | 8.2 [2.3 to 19.6]
  Joint pain: Moderate | 3.4 [1.7 to 6.2] | 2.1 [0.4 to 6.0] | 4.7 [1.9 to 9.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Joint pain: Severe | 1.0 [0.2 to 3.0] | 2.1 [0.4 to 6.0] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.3]
  Antipyretic Medication Use | 29.9 [24.7 to 35.5] | 32.9 [25.2 to 41.2] | 27.0 [20.1 to 34.9] | 5.8 [2.2 to 12.2] | 1.9 [0.0 to 9.9] | 10.2 [3.4 to 22.2]

7. Primary Outcome: Percentage of Participants Reporting Systemic Events and Antipyretic Use Within 7 Days After Vaccination 3
Description: as for outcome 6
Time Frame: Within 7 Days after Vaccination 3
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 285 | 139 | 146 | 104 | 54 | 50
Percentage of participants
  Fever >=38 degrees C | 6.7 [4.1 to 10.2] | 11.5 [6.7 to 18.0] | 2.1 [0.4 to 5.9] | 5.8 [2.1 to 12.1] | 9.3 [3.1 to 20.3] | 2.0 [0.1 to 10.6]
  Fever 38 to <38.5 degrees C | 3.5 [1.7 to 6.4] | 5.0 [2.0 to 10.1] | 2.1 [0.4 to 5.9] | 2.9 [0.6 to 8.2] | 3.7 [0.5 to 12.7] | 2.0 [0.1 to 10.6]
  Fever 38.5 to <39 degrees C | 1.8 [0.6 to 4.0] | 3.6 [1.2 to 8.2] | 0.0 [0.0 to 2.5] | 1.9 [0.2 to 6.8] | 3.7 [0.5 to 12.7] | 0.0 [0.0 to 7.1]
  Fever 39 to <39.5 degrees C | 1.1 [0.2 to 3.0] | 2.2 [0.4 to 6.2] | 0.0 [0.0 to 2.5] | 1.0 [0.0 to 5.2] | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 7.1]
  Fever 39.5 to 40 degrees C | 0.4 [0.0 to 1.9] | 0.7 [0.0 to 3.9] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]
  Fever >40 degrees C | 0.0 [0.0 to 1.3] | 0.0 [0.0 to 2.6] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]
  Vomiting: Any | 3.2 [1.5 to 5.9] | 4.3 [1.6 to 9.2] | 2.1 [0.4 to 5.9] | 3.8 [1.1 to 9.6] | 5.6 [1.2 to 15.4] | 2.0 [0.1 to 10.6]
  Vomiting: Mild | 2.1 [0.8 to 4.5] | 2.9 [0.8 to 7.2] | 1.4 [0.2 to 4.9] | 1.9 [0.2 to 6.8] | 3.7 [0.5 to 12.7] | 0.0 [0.0 to 7.1]
  Vomiting: Moderate | 1.1 [0.2 to 3.0] | 1.4 [0.2 to 5.1] | 0.7 [0.0 to 3.8] | 1.9 [0.2 to 6.8] | 1.9 [0.0 to 9.9] | 2.0 [0.1 to 10.6]
  Vomiting: Severe | 0.0 [0.0 to 1.3] | 0.0 [0.0 to 2.6] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]
  Diarrhea: Any | 6.3 [3.8 to 9.8] | 6.5 [3.0 to 11.9] | 6.2 [2.9 to 11.4] | 2.9 [0.6 to 8.2] | 3.7 [0.5 to 12.7] | 2.0 [0.1 to 10.6]
  Diarrhea: Mild | 5.3 [3.0 to 8.5] | 5.8 [2.5 to 11.0] | 4.8 [1.9 to 9.6] | 2.9 [0.6 to 8.2] | 3.7 [0.5 to 12.7] | 2.0 [0.1 to 10.6]
  Diarrhea: Moderate | 0.7 [0.1 to 2.5] | 0.7 [0.0 to 3.9] | 0.7 [0.0 to 3.8] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]
  Diarrhea: Severe | 0.4 [0.0 to 1.9] | 0.0 [0.0 to 2.6] | 0.7 [0.0 to 3.8] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]
  Headache: Any | 14.0 [10.2 to 18.6] | 7.2 [3.5 to 12.8] | 20.5 [14.3 to 28.0] | 6.7 [2.7 to 13.4] | 1.9 [0.0 to 9.9] | 12.0 [4.5 to 24.3]
  Headache: Mild | 10.5 [7.2 to 14.7] | 5.8 [2.5 to 11.0] | 15.1 [9.7 to 21.9] | 3.8 [1.1 to 9.6] | 0.0 [0.0 to 6.6] | 8.0 [2.2 to 19.2]
  Headache: Moderate | 3.5 [1.7 to 6.4] | 1.4 [0.2 to 5.1] | 5.5 [2.4 to 10.5] | 2.9 [0.6 to 8.2] | 1.9 [0.0 to 9.9] | 4.0 [0.5 to 13.7]
  Headache: Severe | 0.0 [0.0 to 1.3] | 0.0 [0.0 to 2.6] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]
  Fatigue: Any | 33.3 [27.9 to 39.1] | 36.0 [28.0 to 44.5] | 30.8 [23.5 to 39.0] | 17.3 [10.6 to 26.0] | 18.5 [9.3 to 31.4] | 16.0 [7.2 to 29.1]
  Fatigue: Mild | 18.2 [13.9 to 23.2] | 16.5 [10.8 to 23.8] | 19.9 [13.7 to 27.3] | 11.5 [6.1 to 19.3] | 11.1 [4.2 to 22.6] | 12.0 [4.5 to 24.3]
  Fatigue: Moderate | 14.0 [10.2 to 18.6] | 18.0 [12.0 to 25.4] | 10.3 [5.9 to 16.4] | 5.8 [2.1 to 12.1] | 7.4 [2.1 to 17.9] | 4.0 [0.5 to 13.7]
  Fatigue: Severe | 1.1 [0.2 to 3.0] | 1.4 [0.2 to 5.1] | 0.7 [0.0 to 3.8] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]
  Muscle pain: Any | 12.3 [8.7 to 16.7] | 12.9 [7.9 to 19.7] | 11.6 [6.9 to 18.0] | 4.8 [1.6 to 10.9] | 5.6 [1.2 to 15.4] | 4.0 [0.5 to 13.7]
  Muscle pain: Mild | 6.3 [3.8 to 9.8] | 7.2 [3.5 to 12.8] | 5.5 [2.4 to 10.5] | 2.9 [0.6 to 8.2] | 1.9 [0.0 to 9.9] | 4.0 [0.5 to 13.7]
  Muscle pain: Moderate | 5.6 [3.2 to 9.0] | 5.0 [2.0 to 10.1] | 6.2 [2.9 to 11.4] | 1.9 [0.2 to 6.8] | 3.7 [0.5 to 12.7] | 0.0 [0.0 to 7.1]
  Muscle pain: Severe | 0.4 [0.0 to 1.9] | 0.7 [0.0 to 3.9] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]
  Joint pain: Any | 7.4 [4.6 to 11.0] | 7.2 [3.5 to 12.8] | 7.5 [3.8 to 13.1] | 2.9 [0.6 to 8.2] | 0.0 [0.0 to 6.6] | 6.0 [1.3 to 16.5]
  Joint pain: Mild | 3.9 [1.9 to 6.8] | 2.9 [0.8 to 7.2] | 4.8 [1.9 to 9.6] | 2.9 [0.6 to 8.2] | 0.0 [0.0 to 6.6] | 6.0 [1.3 to 16.5]
  Joint pain: Moderate | 3.2 [1.5 to 5.9] | 3.6 [1.2 to 8.2] | 2.7 [0.8 to 6.9] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]
  Joint pain: Severe | 0.4 [0.0 to 1.9] | 0.7 [0.0 to 3.9] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]
  Antipyretic Medication Use | 26.3 [21.3 to 31.8] | 25.2 [18.2 to 33.2] | 27.4 [20.3 to 35.4] | 10.6 [5.4 to 18.1] | 13.0 [5.4 to 24.9] | 8.0 [2.2 to 19.2]

8. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After Vaccination 1
Description: SAE was an adverse event (AE) resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; lack of efficacy in an approved indication. An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship.
Time Frame: Within 30 Days after Vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 0.3 [0.0 to 1.9] | 0.7 [0.0 to 3.8] | 0.0 [0.0 to 2.4] | 0.9 [0.0 to 5.1] | 1.8 [0.0 to 9.7] | 0.0 [0.0 to 7.0]

9. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After Vaccination 2
Description: SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; lack of efficacy in an approved indication. An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship.
Time Frame: Within 30 Days after Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 291 | 143 | 148 | 104 | 54 | 50
Percentage of participants | 0.7 [0.1 to 2.5] | 1.4 [0.2 to 5.0] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]

10. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After Vaccination 3
Description: as for outcome 9
Time Frame: Within 30 Days after Vaccination 3
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 287 | 140 | 147 | 104 | 54 | 50
Percentage of participants | 0.0 [0.0 to 1.3] | 0.0 [0.0 to 2.6] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]

11. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After Any Vaccination
Description: as for outcome 9
Time Frame: Within 30 Days after any vaccination
Population: Safety population: all participants who received at least 1 dose of the investigational product (rLP2086 or HAV/saline) and had safety data available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 1.0 [0.2 to 3.0] | 2.1 [0.4 to 5.9] | 0.0 [0.0 to 2.4] | 0.9 [0.0 to 5.1] | 1.8 [0.0 to 9.7] | 0.0 [0.0 to 7.0]

12. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) During the Vaccination Phase
Description: as for outcome 9
Time Frame: From the Vaccination 1 up to 1 month after Vaccination 3
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 1.4 [0.4 to 3.4] | 2.1 [0.4 to 5.9] | 0.7 [0.0 to 3.7] | 0.9 [0.0 to 5.1] | 1.8 [0.0 to 9.7] | 0.0 [0.0 to 7.0]

13. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) During the Follow-up Phase
Description: as for outcome 9
Time Frame: From 1 month after Vaccination 3 up to 6 months after Vaccination 3
Population: Safety population: all participants who had at least 1 dose of investigational product (rLP2086 or HAV/saline) and had safety data available from after post third-vaccination blood draw to 6 months after last study vaccination. Here "N" signifies number of participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 284 | 137 | 147 | 104 | 54 | 50
Percentage of participants | 0.4 [0.0 to 1.9] | 0.0 [0.0 to 2.7] | 0.7 [0.0 to 3.7] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]

14. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Throughout the Study
Description: as for outcome 9
Time Frame: From Vaccination 1 up to 6 months after Vaccination 3
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 1.7 [0.6 to 3.9] | 2.1 [0.4 to 5.9] | 1.3 [0.2 to 4.8] | 0.9 [0.0 to 5.1] | 1.8 [0.0 to 9.7] | 0.0 [0.0 to 7.0]

15. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended Adverse Event (AE) Within 30 Days After Vaccination 1
Description: A medically attended AE was defined as a non-serious AE that resulted in an evaluation at a medical facility.
Time Frame: Within 30 Days after Vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 13.3 [9.6 to 17.7] | 18.6 [12.6 to 25.9] | 8.1 [4.2 to 13.6] | 13.2 [7.4 to 21.2] | 16.4 [7.8 to 28.8] | 9.8 [3.3 to 21.4]

16. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended Adverse Event (AE) Within 30 Days After Vaccination 2
Description: A medically attended AE was defined as a non-serious AE that resulted in an evaluation at a medical facility.
Time Frame: Within 30 Days after Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 291 | 143 | 148 | 104 | 54 | 50
Percentage of participants | 12.0 [8.5 to 16.3] | 10.5 [6.0 to 16.7] | 13.5 [8.5 to 20.1] | 11.5 [6.1 to 19.3] | 14.8 [6.6 to 27.1] | 8.0 [2.2 to 19.2]

17. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended Adverse Event (AE) Within 30 Days After Vaccination 3
Description: A medically attended AE was defined as a non-serious AE that resulted in an evaluation at a medical facility.
Time Frame: Within 30 Days after Vaccination 3
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 287 | 140 | 147 | 104 | 54 | 50
Percentage of participants | 5.6 [3.2 to 8.9] | 6.4 [3.0 to 11.9] | 4.8 [1.9 to 9.6] | 4.8 [1.6 to 10.9] | 5.6 [1.2 to 15.4] | 4.0 [0.5 to 13.7]

18. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended Adverse Event (AE) Within 30 Days After Any Vaccination
Description: A medically attended AE was defined as a non-serious AE that resulted in an evaluation at a medical facility.
Time Frame: Within 30 Days after any vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 25.9 [20.9 to 31.3] | 29.0 [21.7 to 37.1] | 22.8 [16.3 to 30.4] | 26.4 [18.3 to 35.9] | 30.9 [19.1 to 44.8] | 21.6 [11.3 to 35.3]

19. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended Adverse Event (AE) During the Vaccination Phase
Description: A medically attended AE was defined as a non-serious AE that resulted in an evaluation at a medical facility.
Time Frame: From the Vaccination 1 up to 1 month after the Vaccination 3
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 43.2 [37.5 to 49.1] | 45.5 [37.2 to 54.0] | 40.9 [33.0 to 49.3] | 46.2 [36.5 to 56.2] | 41.8 [28.7 to 55.9] | 51.0 [36.6 to 65.2]

20. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended Adverse Event (AE) During the Follow-up Phase
Description: A medically attended AE was defined as a non-serious AE that resulted in an evaluation at a medical facility.
Time Frame: From 1 month after Vaccination 3 up to 6 months after the Vaccination 3
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 284 | 137 | 147 | 104 | 54 | 50
Percentage of participants | 18.3 [14.0 to 23.3] | 20.4 [14.0 to 28.2] | 16.3 [10.7 to 23.3] | 12.5 [6.8 to 20.4] | 13.0 [5.4 to 24.9] | 12.0 [4.5 to 24.3]

21. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended Adverse Event (AE) Throughout the Study
Description: A medically attended AE was defined as a non-serious AE that resulted in an evaluation at a medical facility.
Time Frame: From the Vaccination 1 up to 6 months after the Vaccination 3
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 48.6 [42.8 to 54.5] | 49.0 [40.6 to 57.4] | 48.3 [40.1 to 56.6] | 50.0 [40.1 to 59.9] | 47.3 [33.7 to 61.2] | 52.9 [38.5 to 67.1]

22. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Within 30 Days After Vaccination 1
Description: A newly diagnosed chronic medical condition was defined as a disease or medical condition that was not identified prior to study start and was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: Within 30 Days after Vaccination 1
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

23. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Within 30 Days After Vaccination 2
Description: as for outcome 22
Time Frame: Within 30 Days after Vaccination 2
Population: Vaccination 2 safety population: all participants who received the second dose of investigational products (rLP2086 or saline) on Month 2 visit.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

24. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Within 30 Days After Vaccination 3
Description: as for outcome 22
Time Frame: Within 30 Days after Vaccination 3
Population: Vaccination 3 safety population: all participants who received the third dose of investigational product (rLP2086 or HAV vaccine) on Month 6 visit.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

25. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Within 30 Days After Any Vaccination
Description: as for outcome 22
Time Frame: Within 30 Days after any vaccination
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

26. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition During the Vaccination Phase
Description: as for outcome 22
Time Frame: From the Vaccination 1 up to 1 month after the Vaccination 3
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

27. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition During the Follow-up Phase
Description: as for outcome 22
Time Frame: From 1 month after Vaccination 3 up to 6 months after the Vaccination 3
Population: Safety population: all participants who had at least 1 dose of investigational product (rLP2086 or HAV/saline) and had safety data available from after post third-vaccination blood draw to 6 months after last study vaccination.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

28. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Throughout the Study
Description: as for outcome 22
Time Frame: From the Vaccination 1 up to 6 months after the Vaccination 3
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

29. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) Within 30 Days After Vaccination 1
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Within 30 Days after Vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 24.1 [19.4 to 29.5] | 29.0 [21.7 to 37.1] | 19.5 [13.4 to 26.7] | 17.9 [11.2 to 26.6] | 21.8 [11.8 to 35.0] | 13.7 [5.7 to 26.3]

30. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) Within 30 Days After Vaccination 2
Description: as for outcome 29
Time Frame: Within 30 Days after Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 291 | 143 | 148 | 104 | 54 | 50
Percentage of participants | 23.0 [18.3 to 28.3] | 19.6 [13.4 to 27.0] | 26.4 [19.5 to 34.2] | 22.1 [14.6 to 31.3] | 27.8 [16.5 to 41.6] | 16.0 [7.2 to 29.1]

31. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) Within 30 Days After Vaccination 3
Description: as for outcome 29
Time Frame: Within 30 Days after Vaccination 3
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 287 | 140 | 147 | 104 | 54 | 50
Percentage of participants | 14.3 [10.5 to 18.9] | 12.9 [7.8 to 19.6] | 15.6 [10.2 to 22.5] | 9.6 [4.7 to 17.0] | 11.1 [4.2 to 22.6] | 8.0 [2.2 to 19.2]

32. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) Within 30 Days After Any Vaccination
Description: as for outcome 29
Time Frame: Within 30 Days after any vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 44.2 [38.5 to 50.1] | 44.8 [36.6 to 53.3] | 43.6 [35.5 to 52.0] | 39.6 [30.3 to 49.6] | 49.1 [35.4 to 62.9] | 29.4 [17.5 to 43.8]

33. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) During the Vaccination Phase
Description: as for outcome 29
Time Frame: From the Vaccination 1 up to 1 month after the Vaccination 3
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 62.6 [56.8 to 68.1] | 62.1 [53.6 to 70.0] | 63.1 [54.8 to 70.8] | 63.2 [53.3 to 72.4] | 63.6 [49.6 to 76.2] | 62.7 [48.1 to 75.9]

34. Primary Outcome: Percentage of Participants With at Least 1 Immediate Adverse Event (AE) After Vaccination 1
Description: Immediate AE was defined as AEs occurring within the first 30 minutes after investigational product administration.
Time Frame: Within 30 minutes after Vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Percentage of participants | 0 [0.0 to 1.2] | 0 [0.0 to 2.5] | 0 [0.0 to 2.4] | 0 [0.0 to 3.4] | 0 [0.0 to 6.5] | 0 [0.0 to 7.0]

35. Primary Outcome: Percentage of Participants With at Least 1 Immediate Adverse Event (AE) After Vaccination 2
Description: Immediate AE was defined as AEs occurring within the first 30 minutes after investigational product administration.
Time Frame: Within 30 minutes after Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 291 | 143 | 148 | 104 | 54 | 50
Percentage of participants | 0 [0.0 to 1.3] | 0 [0.0 to 2.5] | 0 [0.0 to 2.5] | 0 [0.0 to 3.5] | 0 [0.0 to 6.6] | 0 [0.0 to 7.1]

36. Primary Outcome: Percentage of Participants With at Least 1 Immediate Adverse Event (AE) After Vaccination 3
Description: Immediate AE was defined as AEs occurring within the first 30 minutes after investigational product administration.
Time Frame: Within 30 minutes after Vaccination 3
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 287 | 140 | 147 | 104 | 54 | 50
Percentage of participants | 0.3 [0.0 to 1.9] | 0.0 [0.0 to 2.6] | 0.7 [0.0 to 3.7] | 0 [0.0 to 3.5] | 0 [0.0 to 6.6] | 0.0 [0.0 to 7.1]

37. Primary Outcome: Number of Days Participant's Missed School Due to Adverse Event (AE) During the Vaccination Phase
Time Frame: From the Vaccination 1 up to 1 month after the Vaccination 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 294 | 145 | 149 | 106 | 55 | 51
Days | 4.7 (3.1) | 7.0 (3.7) | 4.0 (2.6) | 4.6 (2.6) | 7.3 (2.3) | 4.2 (2.5)

38. Secondary Outcome: Percentage of Participants Aged >=24 Months to <10 Years With hSBA Titer >= LLOQ for Each of the 4 Primary MnB Test Strains 1 Month After Vaccination 3
Description: Percentage of participants achieving hSBA titer >= LLOQ were computed along with corresponding 2-sided 95% CIs. LLOQ was 1:16 for PMB80 (A22) and 1:8 for PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44).
Time Frame: 1 month after Vaccination 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years)
Number analyzed (Participants) | 274 | 97
Percentage of participants
  PMB80 [A22]: number analyzed (Participants) | 135 | 45
  PMB80 [A22] | 87.4 [80.6 to 92.5] | 6.7 [1.4 to 18.3]
  PMB2001 [A56]: number analyzed (Participants) | 139 | 43
  PMB2001 [A56] | 100.0 [97.4 to 100.0] | 20.9 [10.0 to 36.0]
  PMB2948 [B24]: number analyzed (Participants) | 126 | 46
  PMB2948 [B24] | 88.9 [82.1 to 93.8] | 4.3 [0.5 to 14.8]
  PMB2707 [B44]: number analyzed (Participants) | 134 | 50
  PMB2707 [B44] | 79.1 [71.2 to 85.6] | 0.0 [0.0 to 7.1]

39. Secondary Outcome: Percentage of Participants With hSBA Titer >= LLOQ for Each of the 4 Primary MnB Test Strains 1 Month After Vaccination 2 and 6 Months After Vaccination 3
Description: Percentage of participants achieving hSBA titer >= LLOQ were computed along with corresponding 2-sided 95% CIs. LLOQ was 1:16 for PMB80 (A22) and 1:8 for PMB2001 (A56), PMB2948 (B24), and PMB2707 (B44).
Time Frame: 1 month after Vaccination 2 and 6 months after Vaccination 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 274 | 136 | 138 | 97 | 52 | 45
Percentage of participants
  1 Month after Vaccination 2: PMB80 [A22]: number analyzed (Participants) | 130 | 64 | 66 | 45 | 24 | 21
  1 Month after Vaccination 2: PMB80 [A22] | 69.2 [60.5 to 77.0] | 59.4 [46.4 to 71.5] | 78.8 [67.0 to 87.9] | 4.4 [0.5 to 15.1] | 0.0 [0.0 to 14.2] | 9.5 [1.2 to 30.4]
  6 Months after Vaccination 3: PMB80 [A22]: number analyzed (Participants) | 126 | 63 | 63 | 47 | 26 | 21
  6 Months after Vaccination 3: PMB80 [A22] | 32.5 [24.5 to 41.5] | 19.0 [10.2 to 30.9] | 46.0 [33.4 to 59.1] | 8.5 [2.4 to 20.4] | 7.7 [0.9 to 25.1] | 9.5 [1.2 to 30.4]
  1 Month after Vaccination 2: PMB2001 [A56]: number analyzed (Participants) | 133 | 66 | 67 | 43 | 21 | 22
  1 Month after Vaccination 2: PMB2001 [A56] | 100.0 [97.3 to 100.0] | 100.0 [94.6 to 100.0] | 100.0 [94.6 to 100.0] | 16.3 [6.8 to 30.7] | 9.5 [1.2 to 30.4] | 22.7 [7.8 to 45.4]
  6 Months after Vaccination 3: PMB2001 [A56]: number analyzed (Participants) | 131 | 61 | 70 | 46 | 24 | 22
  6 Months after Vaccination 3: PMB2001 [A56] | 82.4 [74.8 to 88.5] | 80.3 [68.2 to 89.4] | 84.3 [73.6 to 91.9] | 19.6 [9.4 to 33.9] | 16.7 [4.7 to 37.4] | 22.7 [7.8 to 45.4]
  1 Month after Vaccination 2: PMB2948 [B24]: number analyzed (Participants) | 128 | 65 | 63 | 45 | 24 | 21
  1 Month after Vaccination 2: PMB2948 [B24] | 57.0 [48.0 to 65.7] | 49.2 [36.6 to 61.9] | 65.1 [52.0 to 76.7] | 8.9 [2.5 to 21.2] | 8.3 [1.0 to 27.0] | 9.5 [1.2 to 30.4]
  6 Months after Vaccination 3: PMB2948 [B24]: number analyzed (Participants) | 129 | 65 | 64 | 47 | 26 | 21
  6 Months after Vaccination 3: PMB2948 [B24] | 15.5 [9.7 to 22.9] | 9.2 [3.5 to 19.0] | 21.9 [12.5 to 34.0] | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 16.1]
  1 Month after Vaccination 2: PMB2707 [B44]: number analyzed (Participants) | 130 | 63 | 67 | 50 | 26 | 24
  1 Month after Vaccination 2: PMB2707 [B44] | 48.5 [39.6 to 57.4] | 57.1 [44.0 to 69.5] | 40.3 [28.5 to 53.0] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  6 Months after Vaccination 3: PMB2707 [B44]: number analyzed (Participants) | 135 | 66 | 69 | 49 | 26 | 23
  6 Months after Vaccination 3: PMB2707 [B44] | 10.4 [5.8 to 16.8] | 12.1 [5.4 to 22.5] | 8.7 [3.3 to 18.0] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.8]

40. Secondary Outcome: Percentage of Participants With Serum Bactericidal Assay Using hSBA Titers >=1:4, >=1:8, >=1:16, >=1:32, >=1:64 and >=1:128 for Each of the 4 Primary Test Strains
Time Frame: Before Vaccination 1, 1 month after Vaccination 2, 1 month after Vaccination 3 and 6 months after Vaccination 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 274 | 136 | 138 | 97 | 52 | 45
Percentage of participants
  Before Vaccination 1: PMB80 [A22] - 1:4: number analyzed (Participants) | 134 | 68 | 66 | 47 | 26 | 21
  Before Vaccination 1: PMB80 [A22] - 1:4 | 12.7 [7.6 to 19.5] | 5.9 [1.6 to 14.4] | 19.7 [10.9 to 31.3] | 6.4 [1.3 to 17.5] | 3.8 [0.1 to 19.6] | 9.5 [1.2 to 30.4]
  Before Vaccination 1: PMB80 [A22] - 1:8: number analyzed (Participants) | 134 | 68 | 66 | 47 | 26 | 21
  Before Vaccination 1: PMB80 [A22] - 1:8 | 11.9 [7.0 to 18.7] | 5.9 [1.6 to 14.4] | 18.2 [9.8 to 29.6] | 6.4 [1.3 to 17.5] | 3.8 [0.1 to 19.6] | 9.5 [1.2 to 30.4]
  Before Vaccination 1: PMB80 [A22] - 1:16: number analyzed (Participants) | 134 | 68 | 66 | 47 | 26 | 21
  Before Vaccination 1: PMB80 [A22] - 1:16 | 9.0 [4.7 to 15.1] | 4.4 [0.9 to 12.4] | 13.6 [6.4 to 24.3] | 6.4 [1.3 to 17.5] | 3.8 [0.1 to 19.6] | 9.5 [1.2 to 30.4]
  Before Vaccination 1: PMB80 [A22] - 1:32: number analyzed (Participants) | 134 | 68 | 66 | 47 | 26 | 21
  Before Vaccination 1: PMB80 [A22] - 1:32 | 3.0 [0.8 to 7.5] | 1.5 [0.0 to 7.9] | 4.5 [0.9 to 12.7] | 4.3 [0.5 to 14.5] | 0.0 [0.0 to 13.2] | 9.5 [1.2 to 30.4]
  Before Vaccination 1: PMB80 [A22] - 1:64: number analyzed (Participants) | 134 | 68 | 66 | 47 | 26 | 21
  Before Vaccination 1: PMB80 [A22] - 1:64 | 0.0 [0.0 to 2.7] | 0.0 [0.0 to 5.3] | 0.0 [0.0 to 5.4] | 2.1 [0.1 to 11.3] | 0.0 [0.0 to 13.2] | 4.8 [0.1 to 23.8]
  Before Vaccination 1: PMB80 [A22] - 1:128: number analyzed (Participants) | 134 | 68 | 66 | 47 | 26 | 21
  Before Vaccination 1: PMB80 [A22] - 1:128 | 0.0 [0.0 to 2.7] | 0.0 [0.0 to 5.3] | 0.0 [0.0 to 5.4] | 2.1 [0.1 to 11.3] | 0.0 [0.0 to 13.2] | 4.8 [0.1 to 23.8]
  1 month after Vaccination 2: PMB80 [A22] - 1:4: number analyzed (Participants) | 130 | 64 | 66 | 45 | 24 | 21
  1 month after Vaccination 2: PMB80 [A22] - 1:4 | 74.6 [66.2 to 81.8] | 65.6 [52.7 to 77.1] | 83.3 [72.1 to 91.4] | 11.1 [3.7 to 24.1] | 8.3 [1.0 to 27.0] | 14.3 [3.0 to 36.3]
  1 month after Vaccination 2: PMB80 [A22] - 1:8: number analyzed (Participants) | 130 | 64 | 66 | 45 | 24 | 21
  1 month after Vaccination 2: PMB80 [A22] - 1:8 | 72.3 [63.8 to 79.8] | 62.5 [49.5 to 74.3] | 81.8 [70.4 to 90.2] | 8.9 [2.5 to 21.2] | 8.3 [1.0 to 27.0] | 9.5 [1.2 to 30.4]
  1 month after Vaccination 2: PMB80 [A22] - 1:32: number analyzed (Participants) | 130 | 64 | 66 | 45 | 24 | 21
  1 month after Vaccination 2: PMB80 [A22] - 1:32 | 41.5 [33.0 to 50.5] | 35.9 [24.3 to 48.9] | 47.0 [34.6 to 59.7] | 4.4 [0.5 to 15.1] | 0.0 [0.0 to 14.2] | 9.5 [1.2 to 30.4]
  1 month after Vaccination 2: PMB80 [A22] - 1:64: number analyzed (Participants) | 130 | 64 | 66 | 45 | 24 | 21
  1 month after Vaccination 2: PMB80 [A22] - 1:64 | 16.9 [10.9 to 24.5] | 14.1 [6.6 to 25.0] | 19.7 [10.9 to 31.3] | 2.2 [0.1 to 11.8] | 0.0 [0.0 to 14.2] | 4.8 [0.1 to 23.8]
  1 month after Vaccination 2: PMB80 [A22] - 1:128: number analyzed (Participants) | 130 | 64 | 66 | 45 | 24 | 21
  1 month after Vaccination 2: PMB80 [A22] - 1:128 | 4.6 [1.7 to 9.8] | 1.6 [0.0 to 8.4] | 7.6 [2.5 to 16.8] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 16.1]
  1 month after Vaccination 3: PMB80 [A22] - 1:4: number analyzed (Participants) | 135 | 68 | 67 | 45 | 25 | 20
  1 month after Vaccination 3: PMB80 [A22] - 1:4 | 92.6 [86.8 to 96.4] | 86.8 [76.4 to 93.8] | 98.5 [92.0 to 100.0] | 11.1 [3.7 to 24.1] | 8.0 [1.0 to 26.0] | 15.0 [3.2 to 37.9]
  T3: PMB80 [A22] - 1:8: number analyzed (Participants) | 135 | 68 | 67 | 45 | 25 | 20
  T3: PMB80 [A22] - 1:8 | 92.6 [86.8 to 96.4] | 86.8 [76.4 to 93.8] | 98.5 [92.0 to 100.0] | 11.1 [3.7 to 24.1] | 8.0 [1.0 to 26.0] | 15.0 [3.2 to 37.9]
  T3: PMB80 [A22] - 1:32: number analyzed (Participants) | 135 | 68 | 67 | 45 | 25 | 20
  T3: PMB80 [A22] - 1:32 | 67.4 [58.8 to 75.2] | 63.2 [50.7 to 74.6] | 71.6 [59.3 to 82.0] | 4.4 [0.5 to 15.1] | 4.0 [0.1 to 20.4] | 5.0 [0.1 to 24.9]
  T3: PMB80 [A22] - 1:64: number analyzed (Participants) | 135 | 68 | 67 | 45 | 25 | 20
  T3: PMB80 [A22] - 1:64 | 39.3 [31.0 to 48.0] | 38.2 [26.7 to 50.8] | 40.3 [28.5 to 53.0] | 2.2 [0.1 to 11.8] | 4.0 [0.1 to 20.4] | 0.0 [0.0 to 16.8]
  T3:PMB80 [A22] - 1:128: number analyzed (Participants) | 135 | 68 | 67 | 45 | 25 | 20
  T3:PMB80 [A22] - 1:128 | 15.6 [9.9 to 22.8] | 14.7 [7.3 to 25.4] | 16.4 [8.5 to 27.5] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 13.7] | 0.0 [0.0 to 16.8]
  T4: PMB80 [A22] - 1:4: number analyzed (Participants) | 126 | 63 | 63 | 47 | 26 | 21
  T4: PMB80 [A22] - 1:4 | 40.5 [31.8 to 49.6] | 25.4 [15.3 to 37.9] | 55.6 [42.5 to 68.1] | 10.6 [3.5 to 23.1] | 11.5 [2.4 to 30.2] | 9.5 [1.2 to 30.4]
  T4: PMB80 [A22] - 1:8: number analyzed (Participants) | 126 | 63 | 63 | 47 | 26 | 21
  T4: PMB80 [A22] - 1:8 | 38.9 [30.3 to 48.0] | 22.2 [12.7 to 34.5] | 55.6 [42.5 to 68.1] | 8.5 [2.4 to 20.4] | 7.7 [0.9 to 25.1] | 9.5 [1.2 to 30.4]
  T4: PMB80 [A22] - 1:32: number analyzed (Participants) | 126 | 63 | 63 | 47 | 26 | 21
  T4: PMB80 [A22] - 1:32 | 19.8 [13.3 to 27.9] | 14.3 [6.7 to 25.4] | 25.4 [15.3 to 37.9] | 2.1 [0.1 to 11.3] | 0.0 [0.0 to 13.2] | 4.8 [0.1 to 23.8]
  T4: PMB80 [A22] - 1:64: number analyzed (Participants) | 126 | 63 | 63 | 47 | 26 | 21
  T4: PMB80 [A22] - 1:64 | 7.9 [3.9 to 14.1] | 4.8 [1.0 to 13.3] | 11.1 [4.6 to 21.6] | 2.1 [0.1 to 11.3] | 0.0 [0.0 to 13.2] | 4.8 [0.1 to 23.8]
  T4: PMB80 [A22] - 1:128: number analyzed (Participants) | 126 | 63 | 63 | 47 | 26 | 21
  T4: PMB80 [A22] - 1:128 | 2.4 [0.5 to 6.8] | 4.8 [1.0 to 13.3] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 16.1]
  T1: PMB2001 [A56] - 1:4: number analyzed (Participants) | 132 | 67 | 65 | 47 | 24 | 23
  T1: PMB2001 [A56] - 1:4 | 10.6 [5.9 to 17.2] | 3.0 [0.4 to 10.4] | 18.5 [9.9 to 30.0] | 19.1 [9.1 to 33.3] | 16.7 [4.7 to 37.4] | 21.7 [7.5 to 43.7]
  T1: PMB2001 [A56] - 1:8: number analyzed (Participants) | 132 | 67 | 65 | 47 | 24 | 23
  T1: PMB2001 [A56] - 1:8 | 8.3 [4.2 to 14.4] | 1.5 [0.0 to 8.0] | 15.4 [7.6 to 26.5] | 14.9 [6.2 to 28.3] | 8.3 [1.0 to 27.0] | 21.7 [7.5 to 43.7]
  T1: PMB2001 [A56] - 1:16: number analyzed (Participants) | 132 | 67 | 65 | 47 | 24 | 23
  T1: PMB2001 [A56] - 1:16 | 8.3 [4.2 to 14.4] | 1.5 [0.0 to 8.0] | 15.4 [7.6 to 26.5] | 14.9 [6.2 to 28.3] | 8.3 [1.0 to 27.0] | 21.7 [7.5 to 43.7]
  T1: PMB2001 [A56] - 1:32: number analyzed (Participants) | 132 | 67 | 65 | 47 | 24 | 23
  T1: PMB2001 [A56] - 1:32 | 6.8 [3.2 to 12.5] | 0.0 [0.0 to 5.4] | 13.8 [6.5 to 24.7] | 12.8 [4.8 to 25.7] | 8.3 [1.0 to 27.0] | 17.4 [5.0 to 38.8]
  T1: PMB2001 [A56] - 1:64: number analyzed (Participants) | 132 | 67 | 65 | 47 | 24 | 23
  T1: PMB2001 [A56] - 1:64 | 3.8 [1.2 to 8.6] | 0.0 [0.0 to 5.4] | 7.7 [2.5 to 17.0] | 6.4 [1.3 to 17.5] | 4.2 [0.1 to 21.1] | 8.7 [1.1 to 28.0]
  T1: PMB2001 [A56] -1:128: number analyzed (Participants) | 132 | 67 | 65 | 47 | 24 | 23
  T1: PMB2001 [A56] -1:128 | 0.8 [0.0 to 4.1] | 0.0 [0.0 to 5.4] | 1.5 [0.0 to 8.3] | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 14.8]
  T2: PMB2001 [A56] - 1:4: number analyzed (Participants) | 133 | 66 | 67 | 43 | 21 | 22
  T2: PMB2001 [A56] - 1:4 | 100.0 [97.3 to 100.0] | 100.0 [94.6 to 100.0] | 100.0 [94.6 to 100.0] | 16.3 [6.8 to 30.7] | 9.5 [1.2 to 30.4] | 22.7 [7.8 to 45.4]
  T2: PMB2001 [A56] - 1:16: number analyzed (Participants) | 133 | 66 | 67 | 43 | 21 | 22
  T2: PMB2001 [A56] - 1:16 | 99.2 [95.9 to 100.0] | 100.0 [94.6 to 100.0] | 98.5 [92.0 to 100.0] | 16.3 [6.8 to 30.7] | 9.5 [1.2 to 30.4] | 22.7 [7.8 to 45.4]
  T2: PMB2001 [A56] - 1:32: number analyzed (Participants) | 133 | 66 | 67 | 43 | 21 | 22
  T2: PMB2001 [A56] - 1:32 | 94.7 [89.5 to 97.9] | 97.0 [89.5 to 99.6] | 92.5 [83.4 to 97.5] | 11.6 [3.9 to 25.1] | 9.5 [1.2 to 30.4] | 13.6 [2.9 to 34.9]
  T2: PMB2001 [A56] - 1:64: number analyzed (Participants) | 133 | 66 | 67 | 43 | 21 | 22
  T2: PMB2001 [A56] - 1:64 | 81.2 [73.5 to 87.5] | 80.3 [68.7 to 89.1] | 82.1 [70.8 to 90.4] | 7.0 [1.5 to 19.1] | 4.8 [0.1 to 23.8] | 9.1 [1.1 to 29.2]
  T2: PMB2001 [A56] - 1:128: number analyzed (Participants) | 133 | 66 | 67 | 43 | 21 | 22
  T2: PMB2001 [A56] - 1:128 | 54.1 [45.3 to 62.8] | 62.1 [49.3 to 73.8] | 46.3 [34.0 to 58.9] | 2.3 [0.1 to 12.3] | 0.0 [0.0 to 16.1] | 4.5 [0.1 to 22.8]
  T3: PMB2001 [A56] - 1:4: number analyzed (Participants) | 139 | 68 | 71 | 43 | 24 | 19
  T3: PMB2001 [A56] - 1:4 | 100.0 [97.4 to 100.0] | 100.0 [94.7 to 100.0] | 100.0 [94.9 to 100.0] | 23.3 [11.8 to 38.6] | 4.2 [0.1 to 21.1] | 47.4 [24.4 to 71.1]
  T3: PMB2001 [A56] - 1:16: number analyzed (Participants) | 139 | 68 | 71 | 43 | 24 | 19
  T3: PMB2001 [A56] - 1:16 | 100.0 [97.4 to 100.0] | 100.0 [94.7 to 100.0] | 100.0 [94.9 to 100.0] | 20.9 [10.0 to 36.0] | 4.2 [0.1 to 21.1] | 42.1 [20.3 to 66.5]
  T3: PMB2001 [A56] - 1:32: number analyzed (Participants) | 139 | 68 | 71 | 43 | 24 | 19
  T3: PMB2001 [A56] - 1:32 | 98.6 [94.9 to 99.8] | 97.1 [89.8 to 99.6] | 100.0 [94.9 to 100.0] | 11.6 [3.9 to 25.1] | 4.2 [0.1 to 21.1] | 21.1 [6.1 to 45.6]
  T3: PMB2001 [A56] - 1:64: number analyzed (Participants) | 139 | 68 | 71 | 43 | 24 | 19
  T3: PMB2001 [A56] - 1:64 | 93.5 [88.1 to 97.0] | 92.6 [83.7 to 97.6] | 94.4 [86.2 to 98.4] | 4.7 [0.6 to 15.8] | 4.2 [0.1 to 21.1] | 5.3 [0.1 to 26.0]
  T3: PMB2001 [A56] - 1:128: number analyzed (Participants) | 139 | 68 | 71 | 43 | 24 | 19
  T3: PMB2001 [A56] - 1:128 | 77.0 [69.1 to 83.7] | 76.5 [64.6 to 85.9] | 77.5 [66.0 to 86.5] | 0.0 [0.0 to 8.2] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 17.6]
  T4: PMB2001 [A56] - 1:4: number analyzed (Participants) | 131 | 61 | 70 | 46 | 24 | 22
  T4: PMB2001 [A56] - 1:4 | 84.0 [76.5 to 89.8] | 82.0 [70.0 to 90.6] | 85.7 [75.3 to 92.9] | 21.7 [10.9 to 36.4] | 20.8 [7.1 to 42.2] | 22.7 [7.8 to 45.4]
  T4: PMB2001 [A56] - 1:16: number analyzed (Participants) | 131 | 61 | 70 | 46 | 24 | 22
  T4: PMB2001 [A56] - 1:16 | 80.2 [72.3 to 86.6] | 77.0 [64.5 to 86.8] | 82.9 [72.0 to 90.8] | 19.6 [9.4 to 33.9] | 16.7 [4.7 to 37.4] | 22.7 [7.8 to 45.4]
  T4: PMB2001 [A56] - 1:32: number analyzed (Participants) | 131 | 61 | 70 | 46 | 24 | 22
  T4: PMB2001 [A56] - 1:32 | 65.6 [56.9 to 73.7] | 59.0 [45.7 to 71.4] | 71.4 [59.4 to 81.6] | 13.0 [4.9 to 26.3] | 16.7 [4.7 to 37.4] | 9.1 [1.1 to 29.2]
  T4: PMB2001 [A56] - 1:64: number analyzed (Participants) | 131 | 61 | 70 | 46 | 24 | 22
  T4: PMB2001 [A56] - 1:64 | 44.3 [35.6 to 53.2] | 39.3 [27.1 to 52.7] | 48.6 [36.4 to 60.8] | 6.5 [1.4 to 17.9] | 8.3 [1.0 to 27.0] | 4.5 [0.1 to 22.8]
  T4: PMB2001 [A56] - 1:128: number analyzed (Participants) | 131 | 61 | 70 | 46 | 24 | 22
  T4: PMB2001 [A56] - 1:128 | 19.1 [12.7 to 26.9] | 16.4 [8.2 to 28.1] | 21.4 [12.5 to 32.9] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  T1: PMB2948 [B24] - 1:4: number analyzed (Participants) | 134 | 67 | 67 | 47 | 26 | 21
  T1: PMB2948 [B24] - 1:4 | 6.7 [3.1 to 12.4] | 4.5 [0.9 to 12.5] | 9.0 [3.4 to 18.5] | 4.3 [0.5 to 14.5] | 3.8 [0.1 to 19.6] | 4.8 [0.1 to 23.8]
  T1: PMB2948 [B24] - 1:8: number analyzed (Participants) | 134 | 67 | 67 | 47 | 26 | 21
  T1: PMB2948 [B24] - 1:8 | 5.2 [2.1 to 10.5] | 3.0 [0.4 to 10.4] | 7.5 [2.5 to 16.6] | 4.3 [0.5 to 14.5] | 3.8 [0.1 to 19.6] | 4.8 [0.1 to 23.8]
  T1: PMB2948 [B24] - 1:16: number analyzed (Participants) | 134 | 67 | 67 | 47 | 26 | 21
  T1: PMB2948 [B24] - 1:16 | 4.5 [1.7 to 9.5] | 3.0 [0.4 to 10.4] | 6.0 [1.7 to 14.6] | 4.3 [0.5 to 14.3] | 3.8 [0.1 to 19.6] | 4.8 [0.1 to 23.8]
  T1: PMB2948 [B24] - 1:32: number analyzed (Participants) | 134 | 67 | 67 | 47 | 26 | 21
  T1: PMB2948 [B24] - 1:32 | 3.0 [0.8 to 7.5] | 1.5 [0.0 to 8.0] | 4.5 [0.9 to 12.5] | 4.3 [0.5 to 14.3] | 3.8 [0.1 to 19.6] | 4.8 [0.1 to 23.8]
  T1: PMB2948 [B24] - 1:64: number analyzed (Participants) | 134 | 67 | 67 | 47 | 26 | 21
  T1: PMB2948 [B24] - 1:64 | 1.5 [0.2 to 5.3] | 1.5 [0.0 to 8.0] | 1.5 [0.0 to 8.0] | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 16.1]
  T1: PMB2948 [B24] - 1:128: number analyzed (Participants) | 134 | 67 | 67 | 47 | 26 | 21
  T1: PMB2948 [B24] - 1:128 | 0.7 [0.0 to 4.1] | 1.5 [0.0 to 8.0] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 16.1]
  T2: PMB2948 [B24] - 1:4: number analyzed (Participants) | 128 | 65 | 63 | 45 | 24 | 21
  T2: PMB2948 [B24] - 1:4 | 60.9 [51.9 to 69.4] | 53.8 [41.0 to 66.3] | 68.3 [55.3 to 79.4] | 8.9 [2.5 to 21.2] | 8.3 [1.1 to 27.0] | 9.5 [1.2 to 30.4]
  T2: PMB2948 [B24] - 1:16: number analyzed (Participants) | 128 | 65 | 63 | 45 | 24 | 21
  T2: PMB2948 [B24] - 1:16 | 50.8 [41.8 to 59.7] | 43.1 [30.8 to 56.0] | 58.7 [45.6 to 71.0] | 8.9 [2.5 to 21.2] | 8.3 [1.0 to 27.0] | 9.5 [1.2 to 30.4]
  T2: PMB2948 [B24] - 1:32: number analyzed (Participants) | 128 | 65 | 63 | 45 | 24 | 21
  T2: PMB2948 [B24] - 1:32 | 22.7 [15.7 to 30.9] | 15.4 [7.6 to 26.5] | 30.2 [19.2 to 43.0] | 4.4 [0.5 to 15.1] | 4.2 [0.1 to 21.1] | 4.8 [0.1 to 23.8]
  T2: PMB2948 [B24] - 1:64: number analyzed (Participants) | 128 | 65 | 63 | 45 | 24 | 21
  T2: PMB2948 [B24] - 1:64 | 9.4 [4.9 to 15.8] | 3.1 [0.4 to 10.7] | 15.9 [7.9 to 27.3] | 4.4 [0.5 to 15.1] | 4.2 [0.1 to 21.1] | 4.8 [0.1 to 23.8]
  T2: PMB2948 [B24] - 1:128: number analyzed (Participants) | 128 | 65 | 63 | 45 | 24 | 21
  T2: PMB2948 [B24] - 1:128 | 4.7 [1.7 to 9.9] | 1.5 [0.0 to 8.3] | 7.9 [2.6 to 17.6] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 16.1]
  T3: PMB2948 [B24] - 1:4: number analyzed (Participants) | 126 | 63 | 63 | 46 | 26 | 20
  T3: PMB2948 [B24] - 1:4 | 92.9 [86.9 to 96.7] | 90.5 [80.4 to 96.4] | 95.2 [86.7 to 99.0] | 6.5 [1.4 to 17.9] | 11.5 [2.4 to 30.2] | 0.0 [0.0 to 16.8]
  T3: PMB2948 [B24] - 1:16: number analyzed (Participants) | 126 | 63 | 63 | 46 | 26 | 20
  T3: PMB2948 [B24] - 1:16 | 84.9 [77.5 to 90.7] | 81.0 [69.1 to 89.8] | 88.9 [78.4 to 95.4] | 4.3 [0.5 to 14.8] | 7.7 [0.9 to 25.1] | 0.0 [0.0 to 16.8]
  T3: PMB2948 [B24] - 1:32: number analyzed (Participants) | 126 | 63 | 63 | 46 | 26 | 20
  T3: PMB2948 [B24] - 1:32 | 46.8 [37.9 to 55.9] | 38.1 [26.1 to 51.2] | 55.6 [42.5 to 68.1] | 2.2 [0.1 to 11.5] | 3.8 [0.1 to 19.6] | 0.0 [0.0 to 16.8]
  T3: PMB2948 [B24] - 1:64: number analyzed (Participants) | 126 | 63 | 63 | 46 | 26 | 20
  T3: PMB2948 [B24] - 1:64 | 18.3 [11.9 to 26.1] | 9.5 [3.6 to 19.6] | 27.0 [16.6 to 39.7] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 16.8]
  T3: PMB2948 [B24] - 1:128: number analyzed (Participants) | 126 | 63 | 63 | 46 | 26 | 20
  T3: PMB2948 [B24] - 1:128 | 7.1 [3.3 to 13.1] | 4.8 [1.0 to 13.3] | 9.5 [3.6 to 19.6] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 16.8]
  T4: PMB2948 [B24] - 1:4: number analyzed (Participants) | 129 | 65 | 64 | 47 | 26 | 21
  T4: PMB2948 [B24] - 1:4 | 20.2 [13.6 to 28.1] | 13.8 [6.5 to 24.7] | 26.6 [16.3 to 39.1] | 2.1 [0.1 to 11.3] | 0.0 [0.0 to 13.2] | 4.8 [0.1 to 23.8]
  T4: PMB2948 [B24] - 1:16: number analyzed (Participants) | 129 | 65 | 64 | 47 | 26 | 21
  T4: PMB2948 [B24] - 1:16 | 14.7 [9.1 to 22.0] | 9.2 [3.5 to 19.0] | 20.3 [11.3 to 32.2] | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 16.1]
  T4: PMB2948 [B24] - 1:32: number analyzed (Participants) | 129 | 65 | 64 | 47 | 26 | 21
  T4: PMB2948 [B24] - 1:32 | 9.3 [4.9 to 15.7] | 6.2 [1.7 to 15.0] | 12.5 [5.6 to 23.2] | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 16.1]
  T4: PMB2948 [B24] - 1:64: number analyzed (Participants) | 129 | 65 | 64 | 47 | 26 | 21
  T4: PMB2948 [B24] - 1:64 | 4.7 [1.7 to 9.8] | 4.6 [1.0 to 12.9] | 4.7 [1.0 to 13.1] | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 16.1]
  T4: PMB2948 [B24] - 1:128: number analyzed (Participants) | 129 | 65 | 64 | 47 | 26 | 21
  T4: PMB2948 [B24] - 1:128 | 3.1 [0.9 to 7.7] | 3.1 [0.4 to 10.7] | 3.1 [0.4 to 10.8] | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 16.1]
  T1: PMB2707 [B44] - 1:4: number analyzed (Participants) | 138 | 67 | 71 | 50 | 26 | 24
  T1: PMB2707 [B44] - 1:4 | 0.7 [0.0 to 4.0] | 0.0 [0.0 to 5.4] | 1.4 [0.0 to 7.6] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T1: PMB2707 [B44] - 1:8: number analyzed (Participants) | 138 | 67 | 71 | 50 | 26 | 24
  T1: PMB2707 [B44] - 1:8 | 0.0 [0.0 to 2.6] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.1] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T1: PMB2707 [B44] - 1:16: number analyzed (Participants) | 138 | 67 | 71 | 50 | 26 | 24
  T1: PMB2707 [B44] - 1:16 | 0.0 [0.0 to 2.6] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.1] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T1: PMB2707 [B44] - 1:32: number analyzed (Participants) | 138 | 67 | 71 | 50 | 26 | 24
  T1: PMB2707 [B44] - 1:32 | 0.0 [0.0 to 2.6] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.1] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T1: PMB2707 [B44] - 1:64: number analyzed (Participants) | 138 | 67 | 71 | 50 | 26 | 24
  T1: PMB2707 [B44] - 1:64 | 0.0 [0.0 to 2.6] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.1] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T1: PMB2707 [B44] - 1:128: number analyzed (Participants) | 138 | 67 | 71 | 50 | 26 | 24
  T1: PMB2707 [B44] - 1:128 | 0.0 [0.0 to 2.6] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.1] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T2: PMB2707 [B44] - 1:4: number analyzed (Participants) | 130 | 63 | 67 | 50 | 26 | 24
  T2: PMB2707 [B44] - 1:4 | 57.7 [48.7 to 63.3] | 66.7 [53.7 to 78.0] | 49.3 [36.8 to 61.8] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T2: PMB2707 [B44] - 1:16: number analyzed (Participants) | 130 | 63 | 67 | 50 | 26 | 24
  T2: PMB2707 [B44] - 1:16 | 43.1 [34.4 to 52.0] | 55.6 [42.5 to 68.1] | 31.3 [20.6 to 43.8] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T2: PMB2707 [B44] - 1:32: number analyzed (Participants) | 130 | 63 | 67 | 50 | 26 | 24
  T2: PMB2707 [B44] - 1:32 | 30.0 [22.3 to 38.7] | 46.0 [33.4 to 59.1] | 14.9 [7.4 to 25.7] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T2: PMB2707 [B44] - 1:64: number analyzed (Participants) | 130 | 63 | 67 | 50 | 26 | 24
  T2: PMB2707 [B44] - 1:64 | 17.7 [11.6 to 25.4] | 27.0 [16.6 to 39.7] | 9.0 [3.4 to 18.5] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T2: PMB2707 [B44] - 1:128: number analyzed (Participants) | 130 | 63 | 67 | 50 | 26 | 24
  T2: PMB2707 [B44] - 1:128 | 10.0 [5.4 to 16.5] | 15.9 [7.9 to 27.3] | 4.5 [0.9 to 12.5] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T3: PMB2707 [B44] - 1:4: number analyzed (Participants) | 134 | 65 | 69 | 50 | 26 | 24
  T3: PMB2707 [B44] - 1:4 | 82.1 [74.5 to 88.2] | 81.5 [70.0 to 90.1] | 82.6 [71.6 to 90.7] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T3: PMB2707 [B44] - 1:16: number analyzed (Participants) | 134 | 65 | 69 | 50 | 26 | 24
  T3: PMB2707 [B44] - 1:16 | 77.6 [69.6 to 84.4] | 80.0 [68.2 to 88.9] | 75.4 [63.5 to 84.9] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T3: PMB2707 [B44] - 1:32: number analyzed (Participants) | 134 | 65 | 69 | 50 | 26 | 24
  T3: PMB2707 [B44] - 1:32 | 65.7 [57.0 to 73.7] | 67.7 [54.9 to 78.8] | 63.8 [51.3 to 75.0] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T3: PMB2707 [B44] - 1:64: number analyzed (Participants) | 134 | 65 | 69 | 50 | 26 | 24
  T3: PMB2707 [B44] - 1:64 | 52.2 [43.4 to 60.9] | 55.4 [42.5 to 67.7] | 49.3 [37.0 to 61.6] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T3: PMB2707 [B44] - 1:128: number analyzed (Participants) | 134 | 65 | 69 | 50 | 26 | 24
  T3: PMB2707 [B44] - 1:128 | 33.6 [25.7 to 42.2] | 36.9 [25.3 to 49.8] | 30.4 [19.9 to 42.7] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.2]
  T4: PMB2707 [B44] - 1:4: number analyzed (Participants) | 135 | 66 | 69 | 49 | 26 | 23
  T4: PMB2707 [B44] - 1:4 | 13.3 [8.1 to 20.3] | 13.6 [6.4 to 24.3] | 13.0 [6.1 to 23.3] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.8]
  T4: PMB2707 [B44] - 1:16: number analyzed (Participants) | 135 | 66 | 69 | 49 | 26 | 23
  T4: PMB2707 [B44] - 1:16 | 8.1 [4.1 to 14.1] | 9.1 [3.4 to 18.7] | 7.2 [2.4 to 16.1] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.8]
  T4: PMB2707 [B44] - 1:32: number analyzed (Participants) | 135 | 66 | 69 | 49 | 26 | 23
  T4: PMB2707 [B44] - 1:32 | 6.7 [3.1 to 12.3] | 6.1 [1.7 to 14.8] | 7.2 [2.4 to 16.1] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.8]
  T4: PMB2707 [B44] - 1:64: number analyzed (Participants) | 135 | 66 | 69 | 49 | 26 | 23
  T4: PMB2707 [B44] - 1:64 | 5.2 [2.1 to 10.4] | 6.1 [1.7 to 14.8] | 4.3 [0.9 to 12.2] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.8]
  T4: PMB2707 [B44] - 1:128: number analyzed (Participants) | 135 | 66 | 69 | 49 | 26 | 23
  T4: PMB2707 [B44] - 1:128 | 3.0 [0.8 to 7.4] | 3.0 [0.4 to 10.5] | 2.9 [0.4 to 10.1] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 14.8]

41. Secondary Outcome: Serum Bactericidal Assay Using Human Complement (hSBA) Geometric Mean Titers (GMTs) for Each of the 4 Primary Test Strains
Time Frame: Before Vaccination 1, 1 month after Vaccination 2, 1 month after Vaccination 3 and 6 months after Vaccination 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 1 Bivalent rLP2086 (>=24 Months to <4 Years) | Group 1 Bivalent rLP2086 (>=4 Years to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <4 Years) | Group 2 HAV/Saline (>=4 Years to <10 Years)
Number analyzed (Participants) | 274 | 136 | 138 | 97 | 52 | 45
titers
  Before Vaccination 1: PMB80 [A22]: number analyzed (Participants) | 134 | 68 | 66 | 47 | 26 | 21
  Before Vaccination 1: PMB80 [A22] | 8.7 [8.3 to 9.1] | 8.3 [7.9 to 8.8] | 9.1 [8.3 to 9.9] | 8.9 [7.8 to 10.1] | 8.2 [7.8 to 8.7] | 9.8 [7.2 to 13.2]
  1 month after Vaccination 2: PMB80 [A22]: number analyzed (Participants) | 130 | 64 | 66 | 45 | 24 | 21
  1 month after Vaccination 2: PMB80 [A22] | 20.1 [17.4 to 23.2] | 17.4 [14.2 to 21.4] | 23.1 [18.9 to 28.3] | 8.6 [7.7 to 9.7] | 8.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 9.4 [7.4 to 12.0]
  1 month after Vaccination 3: PMB80 [A22]: number analyzed (Participants) | 135 | 68 | 67 | 45 | 25 | 20
  1 month after Vaccination 3: PMB80 [A22] | 35.8 [30.5 to 42.2] | 33.7 [26.4 to 42.9] | 38.2 [30.6 to 47.6] | 8.8 [7.8 to 9.8] | 8.7 [7.3 to 10.3] | 8.9 [7.6 to 10.4]
  6 months after Vaccination 3: PMB80 [A22]: number analyzed (Participants) | 126 | 63 | 63 | 47 | 26 | 21
  6 months after Vaccination 3: PMB80 [A22] | 12.4 [10.9 to 14.2] | 10.9 [9.0 to 13.1] | 14.2 [11.8 to 17.0] | 8.7 [7.9 to 9.7] | 8.4 [7.8 to 9.1] | 9.1 [7.4 to 11.3]
  Before Vaccination 1: PMB2001 [A56]: number analyzed (Participants) | 132 | 67 | 65 | 47 | 24 | 23
  Before Vaccination 1: PMB2001 [A56] | 4.9 [4.3 to 5.5] | 4.1 [3.9 to 4.3] | 5.8 [4.6 to 7.3] | 5.6 [4.4 to 7.2] | 4.9 [3.7 to 6.6] | 6.5 [4.3 to 9.8]
  1 month after Vaccination 2: PMB2001 [A56]: number analyzed (Participants) | 133 | 66 | 67 | 43 | 21 | 22
  1 month after Vaccination 2: PMB2001 [A56] | 96.6 [83.0 to 112.5] | 103.8 [84.2 to 127.9] | 90.0 [71.9 to 112.7] | 5.8 [4.4 to 7.6] | 5.0 [3.6 to 7.1] | 6.6 [4.2 to 10.5]
  1 month after Vaccination 3: PMB2001 [A56]: number analyzed (Participants) | 139 | 68 | 71 | 43 | 24 | 19
  1 month after Vaccination 3: PMB2001 [A56] | 183.3 [156.7 to 214.4] | 175.6 [139.1 to 221.6] | 191.0 [153.9 to 237.1] | 6.0 [4.6 to 7.7] | 4.5 [3.5 to 5.7] | 8.6 [5.4 to 13.8]
  6 months after Vaccination 3: PMB2001 [A56]: number analyzed (Participants) | 131 | 61 | 70 | 46 | 24 | 22
  6 months after Vaccination 3: PMB2001 [A56] | 31.3 [25.3 to 38.7] | 27.0 [19.7 to 36.9] | 35.7 [26.6 to 47.8] | 6.0 [4.6 to 7.8] | 6.0 [4.0 to 8.9] | 6.0 [4.2 to 8.7]
  Before Vaccination 1: PMB2948 [B24]: number analyzed (Participants) | 134 | 67 | 67 | 47 | 26 | 21
  Before Vaccination 1: PMB2948 [B24] | 4.5 [4.1 to 4.9] | 4.3 [3.8 to 4.9] | 4.6 [4.0 to 5.2] | 4.4 [3.9 to 4.9] | 4.3 [3.7 to 5.1] | 4.4 [3.6 to 5.4]
  1 month after Vaccination 2: PMB2948 [B24]: number analyzed (Participants) | 128 | 65 | 63 | 45 | 24 | 21
  1 month after Vaccination 2: PMB2948 [B24] | 11.1 [9.2 to 13.5] | 9.1 [7.0 to 11.9] | 13.7 [10.3 to 18.2] | 4.8 [4.0 to 5.8] | 4.8 [3.7 to 6.2] | 4.9 [3.6 to 6.6]
  T3: PMB2948 [B24]: number analyzed (Participants) | 126 | 63 | 63 | 46 | 26 | 20
  T3: PMB2948 [B24] | 22.6 [19.1 to 26.8] | 19.1 [14.9 to 24.5] | 26.8 [21.3 to 33.9] | 4.3 [3.9 to 4.8] | 4.6 [3.8 to 5.6] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means.
  T4: PMB2948 [B24]: number analyzed (Participants) | 129 | 65 | 64 | 47 | 26 | 21
  T4: PMB2948 [B24] | 5.6 [4.8 to 6.5] | 5.1 [4.1 to 6.3] | 6.2 [4.9 to 7.7] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means.
  T1: PMB2707 [B44]: number analyzed (Participants) | 138 | 67 | 71 | 50 | 26 | 24
  T1: PMB2707 [B44] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means.
  T2: PMB2707 [B44]: number analyzed (Participants) | 130 | 63 | 67 | 50 | 26 | 24
  T2: PMB2707 [B44] | 11.7 [9.3 to 14.7] | 17.1 [11.8 to 24.8] | 8.2 [6.3 to 10.6] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means.
  T3: PMB2707 [B44]: number analyzed (Participants) | 134 | 65 | 69 | 50 | 26 | 24
  T3: PMB2707 [B44] | 39.8 [30.6 to 51.6] | 43.6 [29.9 to 63.6] | 36.5 [25.2 to 52.7] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means.
  T4: PMB2707 [B44]: number analyzed (Participants) | 135 | 66 | 69 | 49 | 26 | 23
  T4: PMB2707 [B44] | 5.1 [4.4 to 5.9] | 5.2 [4.2 to 6.4] | 5.0 [4.1 to 6.2] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means.

ADVERSE EVENTS:
Time Frame: AEs/SAEs: Recorded from first vaccination through 6 months after third vaccination. Participants recorded local reactions and systemic events in e-diary within 7 days after first, second and third vaccination.
Description: SAEs and AEs were grouped by system organ class and preferred term. AEs included AEs collected in the e-diary (local and systemic reactions; systematic assessment) and AEs collected on the case report form at each visit (nonsystematic assessment).
Arm/Group | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) | Group 2 HAV/Saline (>=24 Months to <10 Years)
All-Cause Mortality (participants affected / at risk) | 0/294 | 0/106
Serious Adverse Events (participants affected / at risk) | 5/294 | 1/106
Other Adverse Events (participants affected / at risk) | 281/294 | 87/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) (N=294) | Group 2 HAV/Saline (>=24 Months to <10 Years) (N=106)
Bronchitis (Infections and infestations) | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Group 1 Bivalent rLP2086 (>=24 Months to <10 Years) (N=294) | Group 2 HAV/Saline (>=24 Months to <10 Years) (N=106)
Ear pain (Ear and labyrinth disorders) | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (diarrhea) (Gastrointestinal disorders) | 51 | 13
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Teething (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 35 | 13
Vomiting (Gastrointestinal disorders) | 1 | 0
Crying (General disorders) | 0 | 1
Fatigue (General disorders) | 175 | 41
Fatigue (General disorders) | 3 | 0
Injection site erythema (redness) (General disorders) | 177 | 18
Injection site hypersensitivity (General disorders) | 0 | 1
Injection site pain (pain) (General disorders) | 248 | 35
Injection site pain (General disorders) | 4 | 1
Injection site pruritus (General disorders) | 0 | 1
Injection site swelling (swelling) (General disorders) | 137 | 10
Local swelling (General disorders) | 1 | 0
Pyrexia (fever) (General disorders) | 72 | 13
Pyrexia (General disorders) | 16 | 2
Vaccination site pain (General disorders) | 2 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 3 | 0
Bronchitis (Infections and infestations) | 19 | 6
Chronic tonsillitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 9 | 2
Enterobiasis (Infections and infestations) | 0 | 1
Exanthema subitum (Infections and infestations) | 1 | 0
Foot and mouth disease (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 5 | 0
Gastroenteritis (Infections and infestations) | 39 | 10
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 1
Gingivitis (Infections and infestations) | 0 | 1
Herpes dermatitis (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 5 | 0
Infection parasitic (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 6 | 7
Meningitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2
Influenza (Infections and infestations) | 7 | 2
Otitis media acute (Infections and infestations) | 1 | 1
Otitis media viral (Infections and infestations) | 2 | 0
Paronychia (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 33 | 9
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 4
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 12 | 4
Otitis media (Infections and infestations) | 44 | 12
Rhinitis (Infections and infestations) | 4 | 2
Scarlet fever (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin bacterial infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 10 | 3
Upper respiratory tract infection (Infections and infestations) | 59 | 16
Urinary tract infection (Infections and infestations) | 5 | 1
Varicella zoster virus infection (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 7 | 4
Viral upper respiratory tract infection (Infections and infestations) | 31 | 8
Vulvitis (Infections and infestations) | 1/146 | 0/62 — This event is a gender specific event.
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Nasal injury (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 43 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 83 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 98 | 22
Headache (Nervous system disorders) | 6 | 0
Lethargy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Irritability (Psychiatric disorders) | 4 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0/148 | 1/44 — This event is a gender specific event.
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-02-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT02531698/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT02531698/SAP_001.pdf